# 索凡替尼联合卡瑞利珠单抗及mFOLFOX6方案二线治疗晚期胰腺癌的探索性临床研究

课题负责人: 骆卉妍

方案编号: HMPL-012-SPRING-P106

课题研究单位:中山大学附属肿瘤医院

版本号: 2.3 版

版本日期: 2023年12月12日

# 申办者方案签字页

我方已阅读并确认此临床试验方案(方案编号: 版本号: 2.3, 版本日期: 2023年12月12日)。我同意按照中国法律、赫尔辛基宣言、ICH-GCP以及此研究方案履行相关的职责,需经伦理委员会同意后才可实施,除非为保护受试者的安全、权利和利益而必须采取措施。

| 申办单位: 中山大学 | 2附属肿瘤医院 | |
|------------|----------------|-------------|
| 骆卉妍 | | |
| 研究负责人(印刷体) | —<br>研究负责人(签名) | 签字日期(年/月/日) |

# 方案签字页

我将根据中国 GCP 规定认真履行研究者职责,亲自参加或直接指导本临床研究。我已知晓并阅读过该试验药物的临床前研究情况及本项临床试验的研究方案。我同意按照中国法律、赫尔辛基宣言、中国 GCP 以及此研究方案履行相关的职责。我将负责做出与临床相关的医学决定,保证受试者在研究期间出现不良事件时能及时得到适当的治疗,并按照国家有关规定要求记录和报告这些不良事件。我保证将数据真实、准确、完整、及时地记录。

| <b>研究单位:</b> 中山 | 」大学附属肿瘤医院 | <u> </u> |
|-----------------|-----------|----------|
| 骆卉妍 | | |
| 主要研究者(印刷体) | | |

# 方案摘要

| | 走几共日联人上地利亚英长刀 FOLFOX(大安一体沙壳吃知時 |
|---|---|
| 方案名称 | 索凡替尼联合卡瑞利珠单抗及 mFOLFOX6 方案二线治疗晚期胰 |
| | 腺癌的探索性临床研究 |
| | 初步评价索凡替尼联合卡瑞利珠单抗及 mFOLFOX6 方案二线治 |
| 研究目的 | 疗晚期胰腺癌是否有生存获益, 为晚期胰腺癌二线及后线治疗探 |
| | 讨可行性策略 |
| 研究药物 | 索凡替尼、卡瑞利珠单抗 |
| 参研单位 | 中山大学附属肿瘤医院 |
| 主要研究者 | 骆卉妍 |
| | 主要研究终点: |
| | 客观缓解率(ORR) |
| 研究终点 | 次要研究终点: |
| | 疾病控制率(DCR)、缓解持续时间(DOR)、无进展生存期(PFS)、 |
| | 总生存期(OS)、生活质量评分、安全性 |
| 样本量 | 37 例 |
| 研究设计 | 単臂、単中心Ⅱ期临床研究 |
| | 患者必须符合以下所有条件才能入组本研究: |
| | 1. 对本研究已充分了解并自愿签署知情同意书; |
| | 2. 年龄≥18 岁且≤75 岁,男女不限; |
| | 3. 经组织或细胞学确诊的转移性胰腺癌患者; |
| | 4. 既往接受过一线吉西他滨为基础的化疗失败的患者或前期 |
| | 进行新辅助/辅助治疗期间或治疗结束后 6 个月以内出现疾 |
| | 病进展/复发,则认为一线全身化疗失败;新辅助/辅助治疗方 |
| 入选标准 | <br> 案同样为吉西他滨为基础的化疗; |
| | <br> 5. 患者需至少具有一个可测量病灶(RECIST 1.1); |
| | 6. ECOG PS 0-1 分; |
| | <br> 7. 预期生存≥12 周; |
| | 结束后 180 天内采用至少一种经医学认可的避孕措施(如宫 |
| | 内节育器,避孕药或避孕套);且在首次用药前血清 HCG 检 |
| 四节育器, 避孕约或避孕套); 且任自次用约削皿汽<br>查必须为阴性; 而且必须为非哺乳期。 | |
| | 患者若符合以下任何一项标准,将不得进入本研究: |
| 排除标准 | 1. 28 天内参加过其他抗肿瘤药物临床试验; |
| | 1. 20 八門 |

- 2. 既往接受过任何抗 PD-1 抗体、抗 PD-L1 抗体、抗 PD-L2 抗体或抗细胞毒 T 淋巴细胞相关抗原-4(CTLA-4)抗体或作用于 T 细胞协同刺激或检查点通路的任何其它抗体(如 OX40、CD137等)治疗;
- 3. 既往接受过抗血管内皮生长因子/血管内皮生长因子受体 (VEGF/VEGFR) 靶向药物治疗;
- 4. 已知对研究中的任何药物存在过敏者;
- 5. 伴有症状或症状控制时间<2 个月的脑转移;
- 6. 5 年內受试者既往或同时患有其它恶性肿瘤(已治愈的皮肤 基底细胞癌和宫颈原位癌除外);
- 7. 骨髓造血功能不足(14天内未输血状态下):
  - a)绝对中性粒细胞计数 (ANC) <1.5×10 9/L;
  - b)血小板<100×10<sup>9</sup>/L;
  - c) 血红蛋白<8g/dL。
- 8. 肝脏异常:
  - a)无肝转移时,ALT、AST或ALP>2.5×正常值参考范围上限(ULN);肝转移时,ALT、AST或ALP>5\*ULN;
  - b)血清总胆红素>1.5 \*ULN(Gilber 综合症者>3 \*ULN);
  - c)失代偿期肝硬化(Child-Pugh 肝功能评级为 B 或 C

#### 级);

- d)乙肝表面抗原(HBsAg)阳性且乙型肝炎病毒 DNA 拷贝数≥2000IU/mL(HBsAg 阳性且乙型肝炎病毒 DNA 拷贝数 <2000IU/mL 者需至少接受 2 周抗 HBV 治疗才能首次给药);
- e) 丙型肝炎病毒(HCV)抗体阳性且 HCVRNA 检测阳性。
- 9. 肾脏异常:
  - a)血清肌酐>1.5×ULN:
  - b)尿常规提示尿蛋白≥++,且证实 24 小时尿蛋白定量>1.0g;
  - c)肾功能衰竭需要血液透析或腹膜透析;

- d) 既往肾病综合征病史。
- 10. 出血风险:
  - a)凝血功能异常: 部分活化凝血酶原时间(APTT)或凝血酶时间(TT)>1.5×ULN,或国际标准化比值(INR)>1.5(需要抗凝治疗的受试者>2.5);
  - b)患有出血(咯血)、凝血性疾病或正在使用华法林、阿司匹林、低分子肝素及其他抗血小板凝集药物(阿司匹林 ≤100mg/d 预防性用药除外);
  - c)活动性胃肠道出血,表现为在过去3个月内有呕血、便血或黑便,根据内窥镜或结肠镜检查没有消退证据;
  - d)在首次给药前 4 周内,出现任何 CTCAE≥3 级出血或流血事件。
- 11. 心脑血管异常:
  - a)首次给药前 12 个月内有下列任何情况的受试者: ≥II 级心肌缺血或心肌梗死、心律失常, ≥III 级心功能不全, 未控制的心绞痛, 冠状动脉/周围动脉旁路移植手术, 有症状的充血性心力衰竭, 脑血管意外或短暂性脑缺血发作等;
  - b)首次给药前 6 个月内有深静脉血栓或肺栓塞;
  - c)多普勒超声评估的左室射血分数(LVEF) <50%;
  - d)Fridericia 校正后的 QTc 间期(QTcF)平均值(获得至少连续 3 次心电图检测): 男性≥450ms, 女性≥470ms;
  - e)存在药物未能控制的高血压(至少有 2 次测量结果为收缩 压≥150mmHg,舒张压≥100mmHg)。
- 12. 免疫缺陷病史:
  - a)已知人类免疫缺陷病毒(HIV)感染;
  - b)其他获得性、先天性免疫缺陷疾病;
  - c)准备进行或既往接受过器官移植,或首次用药前 60 天内接受过造血干细胞移植,或具有明显的宿主移植反应;

d)需使用免疫抑制剂、或全身、或可吸收的局部激素治疗以 达到免疫抑制目的,并在首次给药前7天内仍需继续使用 的患者(糖皮质激素每日剂量<10mg、泼尼松或其他等疗效 激素除外)。 13. 活动性或未能控制的严重感染: 14. 受试者存在不能口服药物的情况: 15. 研究者认为受试者存在任何临床或实验室检查异常或其他 原因而不适合参加本临床研究。 受试者出现以下的任何一种情况,必须停止治疗,但可继续在研 究中接受监测: 1. 影像学证据表明肿瘤进展: 2. 受试者撤回知情同意,要求退出研究: 终止治疗标 准 3. 无法耐受毒性者; 4. 受试者依从性不佳; 5. 受试者失访; 6. 研究者认为有必要退出研究的情况 所有签署了知情同意书, 筛选合格进入研究的受试者, 均有权随 时退出本研究。 1. 对于只签署了知情同意书, 筛选合格而没有入组的患者, 不作 为脱落病例。 2. 入组后,只要没有完成一个周期的试验无法进行有效性评价 者,均为脱落病例。但是由于以下原因除外: 脱落标准 (1) 入组后因为疾病进展并且有明确的医学证据的,不视为脱 落,但是必须提供影像学证据; (2) 因为受试者怀孕或者毒性不可耐受出组者,也不得视为脱 落; (3) 研究者从受试者的最大利益出发判定应终止治疗; (4) 入组后死亡。 每 6 周 (±7 天) 评估一次疗效, 用药超过 24 周的患者, 每 12 周 治疗方案 (±7天)进行1次疗效评价。疾病控制(CR+PR+SD)且不良反 应可以耐受的受试者,可持续用药,直到失去临床获益、毒性不

| | 可耐受、疗效评价为进展(PD)或免疫治疗证实的疾病进展 |
|---|---|
| | (iCPD)、研究者认为不适合继续用药时研究结束(以先出现者 |
| | 计)。 |
| | 索凡替尼:索凡替尼推荐日剂量为 250mg,每日一次,连续给药; |
| | 卡瑞利珠单抗: 给药剂量固定为 200mg, 在联合用药期间每 14 |
| | 天给药一次,维持治疗期间每21天给药一次,用药最多满2年 |
| | 后停药; |
| | 化疗方案(mFOLFOX6,奥沙利铂+亚叶酸钙+氟脲嘧啶): 奥沙 |
| | 利铂 85mg/m <sup>2</sup> d1+CF 400mg/m <sup>2</sup> d1+5-FU 400mg/m <sup>2</sup> d1/2400mg/m <sup>2</sup> |
| | <br> 持续静注(civ)46h,每 14 天给药一次,共 8-12 个周期,具体 |
| | 周期数由研究者综合判断。 |
| | 安全性评价:采用 NCI-CTCAE5.0 标准评价药物的不良反应。 |
| | 有效性评价: RECIST1.1/iRECIST。本次研究的疗效评估标准依 |
| 评估标准 | 据 RECIST1.1,同时使用 iRECIST 标准对疗效进行确认。即按 |
| | RECIST1.1 标准判定为疾病进展(PD)的受试者,按 iRECIST |
| | <br> 标准进一步确认,从而决定是否继续用药观察。 |
| | 查阅文献知历史对照 ORR: 胰腺癌二线治疗 ORR 为 6%-15%左 |
| | 右,参考多个二线治疗研究结果并结合临床时间,选择 ORR 为 |
| 样本量 | 10%作为历史数据参考,假设卡瑞利珠单抗联合化疗和靶向的 |
| | ORR 为 25%。单侧检验,取I类错误 0.05,基于 0.80 的功效,使 |
| | 用 PASS 软件计算样本量。考虑脱落率 10%,样本量需放大至 |
| | 33/0.9=36.67,向上取整取 37。 |
| | 预计首例受试者入组时间: 2023 年 9 月 |
| 试验时间 | 预计末例受试者入组时间: 2025 年 9 月 |
| | 预计研究结束时间: 2026年9月 |

# 研究访视流程表

| | 筛选 | 期 | 治疗期(14 天) | 为一个治疗周期)12 | 研究治疗结束 | 随访 | 期 |
|---|---|---|---|---|---|---|---|
| | | | 第一周期 | 第二周期及以后 | | | |
| 阶段 | -28至-1天 | -14 至-1<br>天 | D1 | D1 | 获知或确认受试<br>者终止治疗后 | 末次试验用药后 30<br>天 | 生存期访视 13 |
| 时间窗(天) | | | ±7 | ±7 | ±7 | ±7 | ±7 |
| 一般资料 | | | | | | | |
| 书面知情同意 1 | X | | | | | | |
| 入选/排除标准 | | X | | | | | |
| 人口统计学/既往<br>病史 | X | | | | | | |
| 伴随用药 | | | У | X. | 1 | | |
| 实验室检测 | | | | | | | |
| 血常规2 | | X | X (按需) | X | X | X | |
| 血生化3 | | X | X (按需) | X | X | X | |
| 尿常规 4 | | X | X (按需) | X | X | X | |
| 大便常规 | | X | X (按需) | X | X | | |
| 凝血功能检查5 | | X | X (每2周 | ]期检查1次) | X | | |
| 甲状腺功能 | | X | X (每 2 周 | ]期检查1次) | X | | |
| 妊娠检查6 | | X | | | X | | |
| 病毒学检测 | | | | | | | |
| (HBV, HCV, | X | | | | | | |
| HIV) | | | | | | | |
| 心脏彩超 | X | | | | | | |
| 临床评估/检查 | | | | | | | |
| 身高 7, 体重 | | X | X | X | | | |

研究方案 2.3 版 (版本日期 2023 年 12 月 12 日)

| | 筛选 | 期 | 治疗期(14 天) | 为一个治疗周期)12 | 研究治疗结束 | 随访 | 期 |
|---|---|---|---|---|---|---|---|
| | | | 第一周期 | 第二周期及以后 | | | |
| 阶段 | -28至-1天 | -14 至-1<br>天 | D1 | D1 | 获知或确认受试<br>者终止治疗后 | 末次试验用药后 30<br>天 | 生存期访视 13 |
| 时间窗(天) | | | ±7 | ±7 | ±7 | ±7 | ±7 |
| 生命体征8 | | X | X | X | X | X | |
| ECOG 评分 | | X | X | X | X | X | |
| 体格检查 9 | | X | X | X | X | X | |
| 12 导联心电图 10 | X | | X | X | X | | |
| 不良事件评估 | 自签署知情同意书至末次用药后 30 天 | | | | | | |
| 研究药物给药 | | | | | | | |
| 索凡替尼(每日 | | | X | X | | | |
| 口服) | | | Α | A | | | |
| 疗效评估 | | | | | | | |
| 肿瘤影像学评估 | X | | 每 6 周/12 月 | 周(±7 天)1 次 | X | | |
| 治疗结束后随访 | | | | | | | |
| 生存状态 | | | | | | | X |

注:除表中所列检查项目及时间点外,研究者可随时增加访视及其他检查项目,检查结果填写在 CRF《常规访视外检查》。本研究接收在当地二甲以上医院进行的检查结果,但疗效评估尽量在本中心进行。

- 1. 签署知情同意书应在任何方案规定的操作之前进行。
- 2. 血液学检查:全血计数(绝对值)包括红细胞计数、白细胞及分类计数(中性粒细胞、淋巴细胞、单核细胞、嗜酸性粒细胞和嗜碱性粒细胞)、血小板计数,血红蛋白和红细胞压积,在首次使用研究药物前 14 天内完成。如果受试者没有临床症状和指征,第1周期第1天访视不需要重复检查,从第2周期开始每个周期第1天完成和在安全性随访期进行。有临床指征时,可进行计划外的检查。
- 3. 临床生化包括 ALT、AST、总胆红素、直接胆红素、间接胆红素、BUN(尿素氮)或尿素、Cr(血肌酐)、血糖、钾、钠、氯、钙、磷、镁、总蛋白、白蛋白、LDH(乳酸脱氢酶)、ALP(碱性磷酸酶),肌酸激酶,胰淀粉酶或血淀粉酶,甘油三酯和总胆固醇,在首次使用研究药物前 14 天内完成检查。如果受试者没有临床症状和指征,第 1 周期第 1 天访视不需要重复检查。
- 4. 筛选期尿常规检查显示尿蛋白≥++的受试者,应进行 24 小时尿蛋白定量。如果受试者没有临床症状和指征,第1周期第1天访视不需要重复检查。

- 5. 凝血功能检查包括: INR、APTT、PT、FIB。凝血功能及甲状腺功能(血清游离三碘甲状腺原氨酸 FT3、血清游离甲状腺素 FT4 和促甲状腺激素 TSH)每两周期检测一次。
- 6. 有潜在生育能力的女性首次用药前进行血妊娠检测,且 HCG 结果为阴性。经研究者判断,无潜在生育能力的女性可以不进行该项检测。
- 7. 仅在筛选期检测身高,此后不再重复测量身高。
- 8. 生命体征包括:体温、脉博、呼吸频率和血压。
- 9. 体格检查:主要身体系统的检查(头面部、皮肤系统、淋巴结、眼部、耳鼻喉部、口腔、呼吸系统、心血管系统、腹部、生殖泌尿系统、肌肉骨骼、神经系统和精神状态)。除筛选期体格检查外,试验期间无须在 CRF 中记录完整的体格检查结果,只需记录异常情况(仍需进行全面的体格检查)。
- 10. 心电图检查显著异常者,研究者根据受试者情况选择加查心脏超声检查。
- 11. 受试者在接受治疗后,每6周(±7天)接受一次肿瘤影像学评估,用药超过24周的患者,每12周(±7天)接受一次影像学评估,直至失去临床获益、毒性不可耐受、疗效评价疾病进展(PD)或免疫治疗证实的疾病进展(iCPD)、研究者认为不适合继续用药研究结束;如怀疑新发病灶可适时检查;本次研究的疗效评估标准依据RECIST1.1,同时使用iRECIST标准对疗效进行确认,即按RECIST1.1标准判定为疾病进展(PD)的受试者,按iRECIST标准进一步确认,从而决定是否继续用药观察。
- 12. 治疗期: 二线治疗阶段,一个治疗周期为14天;二线维持治疗阶段,一个治疗周期为21天。
- 13. 生存随访: 生存访视每 3 个月(±7 天)进行一次,可以接受电话访视。

# 缩略语与术语定义表

本研究方案采用下列缩略语和专业术语。

| 缩略语与专业术语 | 注释 |
|----------|-----------------|
| ATP | 三磷酸腺苷 |
| AST | 天门冬氨酸氨基转移酶 |
| ALT | 丙氨酸氨基转移酶 |
| AE | 不良事件 |
| CI | 置信区间 |
| CA125 | 糖类抗原-125 |
| CR | 临床完全缓解 |
| CRF | 病例报告表 |
| CT | 计算机断层扫描 |
| CTCAE | 不良事件常见术语标准 |
| DNA | 脱氧核糖核酸 |
| DCR | 疾病控制率 |
| EC | 依托泊苷+卡铂 |
| ECG | 心电图 |
| ECOG | 东部肿瘤协作组 |
| EP | 依托泊苷+顺铂 |
| FAS | 全集分析 |
| FF | 氟尿嘧啶类+亚叶酸钙 |
| FGF | 成纤维细胞生长因子 |
| FOLFOX | 奥沙利铂+氟尿嘧啶类+亚叶酸钙 |
| GCP | 药物临床试验质量管理规范 |
| HR | 风险比 |
| ICH | 国际协调会议 |
| ITT | 意向性治疗 |
| KM | Kaplan Meier 曲线 |
| mFOLFOX6 | 可调整 FOLFOX 方案 |

| MRI | 核磁共振成像 |
|--------|--------------------------------|
| NCI | 国家癌症研究所 |
| NYHA | 纽约核心协会 |
| OFF | 奥沙利铂+氟尿嘧啶类+亚叶酸钙 |
| ORR | 客观缓解率 |
| OS | 总生存期 |
| PD | 疾病进展 |
| PDGF | 血小板衍生生长因子 |
| PFS | 无进展生存期 |
| PR | 部分缓解 |
| QT | QT 间期(心电图 Q 波起始至 T 波(非 U 波)结束) |
| RECIST | 实体瘤疗效评价标准 |
| SAE | 严重不良事件 |
| SD | 病情稳定 |
| TKI | 酪氨酸激酶抑制剂 |
| UNL | 正常值上限 |
| VEGF | 血管内皮生长因子 |

# 目录

| 1. | 研究背景 | 2 |
|----|---------------------------|------|
| 1 | 1.1 胰腺癌流行病学及治疗现状 | 2 |
| 1 | 1.2 科学依据 | 3 |
| 1 | 1.3 索凡替尼的临床前研究总结 | 4 |
| 1 | 1.4 索凡替尼 I /Ib/II 期临床研究结果 | 5 |
| 1 | I.5 索凡替尼 III 期临床研究结果 | 6 |
| 2. | 研究目的和终点 | 8 |
| 2 | 2.1 研究目的 | 8 |
| 2 | 2.2 研究终点 | 8 |
| 3. | 研究设计 | 8 |
| 3 | 3.1 总体设计 | 8 |
| 4. | 受试者的选择和退出 | 9 |
| 2 | 4.1 入选标准 | 9 |
| 2 | 1.2 排除标准 | 9 |
| 2 | 4.3 脱落标准 | . 11 |
| 2 | 1.4 受试者终止治疗标准 | . 12 |
| 5. | 研究实施 | . 12 |
| 4 | 5.1 研究药物 | . 12 |
| 4 | 5.2 给药剂量和方法 | . 13 |
| | 5.2.1 给药剂量 | . 13 |
| | 5.2.2 剂量调整 | . 13 |
| 6. | 研究程序 | . 22 |
| 6 | 6.1 筛选评估(-28~0 天) | . 22 |
| 6 | 6.2 治疗期 | . 23 |
| 6 | 6.3 治疗结束/退出研究评估 | . 24 |
| 6 | 6.4 随访期 | . 24 |
| | 6.4.1 安全性随访 | . 24 |
| | 6.4.2 生存随访 | . 24 |
| 7. | 研究评价和程序 | . 24 |
| - | 7.1 基线评估 | . 24 |

| 7.2 安全性评估 | . 24 |
|----------------------------------|------|
| 7.3 有效性评估 | . 25 |
| 8. 不良事件报告 | . 25 |
| 8.1 不良事件定义(AE) | . 25 |
| 8.2 不良事件的记录 | 26 |
| 8.3 不良事件的程度 | 26 |
| 8.4 不良事件与药物的相关性评价 | . 26 |
| 8.5 严重不良事件 (SAE) | . 27 |
| 9. 统计学分析 | . 28 |
| 9.1 样本量确定 | . 28 |
| 9.2 统计方法 | . 29 |
| 9.2.1 有效性分析 | . 29 |
| 9.3.2 安全性分析 | . 30 |
| 10. 数据收集和管理 | 31 |
| 10.1 病例报告表(CRF) | . 31 |
| 10.2 数据管理 | . 31 |
| 11. 伦理道德 | . 31 |
| 11.1 研究者的责任 | . 31 |
| 11.2 伦理委员会 | . 32 |
| 11.3 受试者信息 | . 32 |
| 11.4 知情同意书 | 32 |
| 12. 参考文献列表 | . 34 |
| 13. 附件一: 实体瘤疗效评价标准(RECIST 1.1 版) | . 36 |
| 14. 附件二: ECOG 体力状况计分标准 | . 44 |
| 15. 附件三: 纽约心脏病学会心功能分级(NYHA) | . 45 |
| 16. 附件四. 索凡替尼与伴随用药潜在相互作用的指导原则 | . 46 |

#### 1. 研究背景

#### 1.1 胰腺癌流行病学及治疗现状

胰腺癌被称为癌中之王,是预后最差的常见实体恶性肿瘤之一,具有恶性程度高、预后差的特点,全球总体发病率和死亡率逐年上升,2020年导致全球46.6万例死亡<sup>[1]</sup>,居所有恶性肿瘤第七位。我国胰腺癌死亡率居所有恶性肿瘤第六位,在2020年新发病例达12.5万例,死亡病例达12.2万例。经预测,至2030年胰腺癌将成为全球第二大癌症死因。

胰腺癌主要治疗手段包括手术切除、化疗、放疗和生物治疗等,但治疗效果均不理想,是治疗效果最差的恶性肿瘤之一。5年总生存率(OS)不到10%,在恶性肿瘤中最低<sup>[2]</sup>,预测2030年,胰腺癌死亡率将仅次于肺癌<sup>[3]</sup>。目前手术治疗结合辅助治疗仍然是胰腺癌患者能获得长期生存机会的唯一方法,然而80%以上的晚期胰腺癌患者丧失了手术的可能,积极的行内科治疗尤为重要。局部进展期或合并远处转移的胰腺癌总体治疗效果不佳,中位生存期在6-9个月,建议开展相关临床研究。

2022 年 CSCO 指南推荐转移性胰腺癌患者一线治疗方案,应根据患者体能状态进行选择,对于体能状态良好的患者,可以考虑联合方案,体能状态较差患者选择单药化疗(GEM 或替吉奥单药)或最佳支持治疗。目前对于转移性胰腺癌患者,标准治疗一般采取联合化疗。其中,一线化疗方案目前有 2 个国际公认标准:奥沙利铂+伊立替康+5-FU/亚叶酸(FOLFIRINOX)三药方案和白蛋白紫杉醇+吉西他滨(AG)两药方案,其中 FOLFIRINOX 方案预期有效率为30%,预期生存11-12 个月,AG 方案预期有效率为25%~30%,预期生存8.5-11 个月[4-7]。AG 方案和 FOLFIRINOX 方案可以互为一线二线,即患者一线耐药后可以更换另一种方案继续治疗,对两种方案的回顾性研究显示,使用顺序不影响患者预后[8]。尽管白蛋白结合紫杉醇联合吉西他滨或 FOLFIRINOX 化疗方案已被证明对胰腺癌患者有显著的生存获益,但其进一步的疗效仍存在挑战。

二线治疗方案目前 CSCO 指南推荐体能状态良好的患者接受纳米脂质体伊利替康联合 5-FU/LV; NAPOLI-1 研究为随机对照III期临床研究<sup>[9-10]</sup>,纳米脂质体伊立替康+5-FU/LV 的 mOS 为 6.1 个月,5-FU/LV 为 4.2 个月(HR=0.67,P=0.012),两组差异有统计学意义。NAPOLI-1 研究共纳入亚洲患者 132 例(韩国和中国台湾),亚洲患者的亚组分析结果显示,纳米脂质体伊立替康+5-FU/LV 的 mOS 为 8.9 个月,5-FU/LV 为 3.7 个月(HR = 0.51,P = 0.025)。其他推荐方案还包括:一线使用吉西他滨为基础的方案,二线建议以 5-FU 为基础的方案;一线使用 5-FU 类为基础的方案,二线建议使用吉西他滨为基础的方案;对于术后发生远处转移者,若距离辅助治疗结束时间>6 个月,除选择原方案全身化疗外,也可选择替代性化疗方案;参加临床研究。

mFOLFOX6 方案为氟尿嘧啶和奥沙利铂为基础的化疗方案,不同的用药剂量和顺序已被证明氟尿嘧啶和奥沙利铂为基础的化疗方案二线治疗转移性胰腺癌的有效性。其中 CONKO-003 研究中,OFF 方案的 OS(5.9 个月 vs 3.3 个月)和 PFS(2.9 个月 vs 2.0 个月)都高于 FF 方案[11]。Yoo C 等开展的研究中证实,mFOLFOX6 方案的 ORR(7% vs 0)和主要研究终点 6 个月的 PFS 率(30% vs 27%)略高于 mFOLFIRI.3 外,OS 和 PFS 均不及 mFOLFIRI.3 方案 [12]。此外,SEQUOIA 研究还对 Pegilodecakin(PEG)联合 FOLFOX 与 FOLFOX 方案的疗效进行了对比,结果显示联合治疗组和单纯化疗组疗效相当[13]。

综上,目前针对晚期胰腺癌二线治疗,单一的治疗手段疗效欠佳,免疫联合治疗也未满足晚期胰腺癌患者的治疗需求,仍需探索新的治疗方法。

#### 1.2 科学依据

本项临床研究涉及的索凡替尼是一种小分子激酶抑制剂,对血管内皮细胞生长因子受体 1、2 和 3(vascular endothelial growth factor receptor,VEGFR),成纤维细胞生长因子受体 1(fibroblast growth factor receptor 1, FGFR1)和集落刺激因子 1 受体(colony stimulating factor 1 receptor,CSF-1R)激酶活性显示出强效抑制作用,其半数抑制浓度(IC50)范围为 1~24 nM,是和记黄埔医药(上海)有限公司独家开发的专利产品。近来有研究证实 FGFR 和 CSF-1R 可以诱导肿瘤相关巨噬细胞的增殖和分化,进而介导肿瘤免疫的调节。因此索凡

替尼在抗血管生成,促进血管正常化方面具有良好的效果;同时,可调节 TAM,改善免疫微环境,促进免疫应答,具有提高免疫治疗疗效的作用机制。 索凡替尼目前已被中国国家药品监督管理局(NMPA)批准用于晚期胰腺和非胰腺神经内分泌瘤治疗。获批是分别是基于中国随机、双盲、安慰剂对照的 III 期临床试验 SANET-p 和 SANET-ep 研究<sup>[14,15]</sup>,在 SANET-ep 研究中,索凡替尼可显著延长患者 PFS(9.2 vs 3.8 个月),提高患者 ORR(10% vs 0%),其中 63%的 ep-NET 患者实现肿瘤退缩获益;在 SANET-p 研究中,索凡替尼可显著 延长患者 PFS(10.9 vs 3.7 个月),提高患者 ORR(19.2% vs 1.9%),其中 84%的 p-NET 患者实现肿瘤退缩获益。两项研究最常见的 3 级及以上不良反应均为高血压和蛋白尿,是抗血管生成 TKI 常出现的不良反应,在临床上可管理。

VEGF家族成员在胰腺导管腺癌(PDAC)中过度表达,在 PDAC 的恶性进展中起重要作用,已经发现 VEGFR1 和 VEGFR2 在 PDAC 中过度表达并促进肿瘤进展。VEGFR1 还被发现可诱导上皮-间充质转化(EMT),这一过程使极化上皮细胞呈现间充质和侵袭表型。VEGFR2 可增强 PDAC 细胞的局部侵袭性,以上提示 VEGF 靶向治疗可能阻断 PDAC 细胞的增殖、存活和运动性[16,17]。VEGFR 参与多种血管生成过程,包括血管渗透、内皮细胞增殖、迁移和生存。血管生成对于恶性肿瘤的生长至关重要。抗血管生成类的分子靶向药物在治疗多种恶性肿瘤中取得了良好的效果。VEGF 在超过 90%的胰腺癌中高表达。一项 II 期临床研究显示,舒尼替尼用于转移性胰腺癌的维持治疗可改善预后。

综上,我们设计了索凡替尼联合卡瑞利珠单抗和 mFOLFOX6 方案二线及后线治疗晚期胰腺癌的探索性研究,以期为晚期胰腺癌患者提供一个安全有效,可耐受的选择,延长其生存时间及改善生活质量。

#### 1.3 索凡替尼的临床前研究总结

我们研究了索凡替尼对 67 种激酶的抑制活性,结果显示索凡替尼对 VEGFR-1/2/3、FGFR-1 和 CSF-1R 有很强的抑制作用,半数抑制浓度分别为 2、24、1、

15 和 4nM,对其余激酶的抑制都比较弱,大多数半数抑制浓度都大于 100nM,显示了较好的选择性。

在细胞水平上,索凡替尼对 VEGF 刺激后 VEGFR-2 的磷酸化以及 VEGF 依赖的 HUVEC 细胞增殖均有明显的抑制,半数抑制浓度分别为 3nM 和 16nM;而对 HUVEC 细胞和其他受试人体肿瘤细胞的直接毒性较弱,半数抑制浓度均大于5000nM。在离体器官组织水平,索凡替尼对大鼠主动脉环微血管的形成也有抑制作用,其 IC50 为 192nM。

在体研究显示,索凡替尼可剂量依赖地抑制 VEGF 刺激的肺组织血管 VEGFR-2 磷酸化,血药浓度大于 181ng/ml 可完全抑制 VEGFR-2 磷酸化,20 mg/kg 的抑制作用可持续 4 小时,因此在裸鼠的肿瘤抑制药效学研究中采用一日 2 次给药方式。

在人胃癌 BGC-823、结肠癌 HT-29、非小细胞肺癌 H460 和肾癌 Caki-1 的裸鼠皮下移植瘤模型上,索凡替尼可剂量依赖性地抑制肿瘤生长,最低有效剂量为 20mg/kg,一日 2 次。药代动力学和药效学的相关性研究也表明索凡替尼抑瘤作用随药物暴露量增加而增强。在最敏感的瘤株胃癌 BGC-823,高剂量下大部分动物出现肿瘤体积缩小(较测量起始平均体积缩小 20%)。在受到抑制的肿瘤组织中,索凡替尼剂量依赖地减少血管内皮特异性表面标记 CD31 阳性细胞的面积,提示肿瘤组织中的血管生成得到抑制。

这些研究提示索凡替尼在临床上有望用于治疗多种实体瘤。

#### 1.4 索凡替尼 I /Ib/II 期临床研究结果

I 期剂量递增临床研究中接受索凡替尼治疗的 18 名疗效可评价的神经内分泌瘤受试者中有 8 名受试者获得 PR (44.4%), 其中在 7 名疗效可评价的 PNET 受试者中,有 3 名达到 PR (42.9%)。另外在神经内分泌瘤受试者中进行的 Ib/II 扩展期研究也出现相似的疗效趋势,显示出索凡替尼在晚期 NETs 的初步疗效。

在 2020 美国癌症研究协会 (AACR) 大会上,索凡替尼 (250mg QD) +特瑞普利单抗的 I 期研究纳入了 30 例既往标准治疗无效的晚期实体瘤受试者,在 29 例可评估的受试者中,总体 DCR 为 79.3%,ORR 为 34.5%。特瑞普利单抗与 250mg、200mg、300mg 索凡替尼治疗后受试者的生存均有获益 (DCR: 100% vs

50% vs 75%; ORR: 63.6% vs 16.7% vs16.7%)。初步证实了索凡替尼联合免疫治疗有协同抗肿瘤作用,并且耐受良好。

基于 I 期的良好结果,后续开展了多队列的 II 期单臂,多中心研究,以进一步验证研究索凡替尼联合特瑞普利单抗治疗晚期实体瘤的疗效与安全性。在安全性方面,索凡替尼 I 期剂量递增研究显示索凡替尼安全性和耐受性较好,尽管未达到最大耐受剂量,但索凡替尼 300 mg QD 剂量水平在人体内的药物暴露量已趋于饱和,遂在 350 mg QD 剂量后未再做更高剂量的探索。索凡替尼 300 mg QD 和 350 mg QD 均为临床有效剂量,且在相同的治疗时间窗内比较,300mg QD 剂量组的≥3 级不良反应较少。因此结合临床药物安全性、耐受性、疗效、药代动力学的结果,确定 II 期临床试验的推荐剂量为 300 mg,口服,每天一次,连续用药。

索凡替尼临床 Ib/II 期试验是一项研究索凡替尼治疗 1 级或 2 级晚期神经内分泌瘤有效性及安全性的开放标签的单臂研究。Ia 期临床试验数据显示索凡替尼的药物不良反应与同类 VEGFR 靶向治疗药物相似,未发现新的安全性信息。这些不良反应多为轻到中度,所引起的治疗中断或减量的发生率较低,且经过对症处理均可得到减轻或恢复。研究中最常见的不良反应包括腹泻、高血压、蛋白尿、腹部不适、AST 升高、血白蛋白降低、乏力等,其发生率和严重程度较同类VEGFR 靶向药物相似或略低;同类靶向药物多发的不良反应如手足综合征在索凡替尼治疗过程中不常见,且未观察血栓栓塞等 VEGFR 靶向药物常见的严重不良反应。索凡替尼的耐受性良好,最常见的≥级治疗相关不良事件为高血压(33%),蛋白尿(12%),高尿酸血症(10%),高甘油三酯血症和腹泻(各为6%)和丙氨酸转氨酶升高(5%)。更为重要的是,1 名接受苏尼替尼和依维莫司治疗后疾病进展的受试者均从索凡替尼治疗中获益(3 名部分缓解、9 名病情稳定)。

#### 1.5 索凡替尼 III 期临床研究结果

索凡替尼目前已被中国国家药品监督管理局(NMPA)批准用于晚期胰腺和非胰腺神经内分泌瘤治疗。获批是分别是基于中国随机、双盲、安慰剂对照的 III 期临床试验 SANET-ep 和 SANET-p 研究。两项研究在中期分析时均达到了预先设定的提前终止研究的标准,因此经独立数据审查委员会批准提前终止研究。

2020 年 9 月, SANET-ep 和 SANET-p 两项研究同期全文在线发表于《柳叶刀•肿瘤》(Lancet Oncology)。

SANET-ep 和 SANET-p 研究均由解放军总医院第五医学中心的徐建明教授牵头。其中 SANET-ep 研究共入组 198 例不可切除或转移性、分化良好的非胰腺来源神经内分泌瘤(NET)患者,体力状态良好(ECOG PS 评分 0 或 1),既往最多接受过 2 种系统性治疗方案后进展。以 2:1 的比例分配,索凡替尼组 129 例,安慰剂组 69 例。主要终点为研究者评估的无进展生存期(PFS)。2019 年 9 月的ESMO 大会上,徐建明教授口头报告了该研究的首次结果,索凡替尼组客观缓解率(ORR)达 10.3%,肿瘤退缩率 63%,疾病控制率(DCR)为 86.5%。索凡替尼组和安慰剂组的中位随访时间分别为 13.8 个月和 16.6 个月,研究者评估的中位 PFS 分别为 9.2 个月和 3.8 个月,索凡替尼显著降低疾病进展或死亡风险达67%。

SANET-p 研究是一项随机、双盲、安慰剂对照、多中心Ⅲ期临床试验,入组 人群为处于疾病进展期、无法手术切除的局部晚期或远处转移的低、中级别(G1 或 G2) p-NET 受试者。在该研究中,受试者以 2:1 的比例随机接受每天口服一 次 300 mg 索凡替尼或安慰剂治疗,28 天为一个治疗周期。研究的主要终点为研 究者评估的无进展生存期(PFS)。SANET-p研究中期数据分析截止时(2019年 11 月 11 日 ), 共入组 172 例晚期胰腺 NET 受试者, 随机接受索凡替尼 (113 例) 或安慰剂(59例)治疗。两组受试者基线特征较为均衡,其中中级别(G2)受 试者所占比重较大(索凡替尼组占87.6%,安慰剂组占84.7%)。结果显示,与安 慰剂相比,索凡替尼能够显著延长研究者评估的 PFS,索凡替尼和安慰剂组分别 为10.9个月和3.7个月,风险比(HR)为0.491[95%可信区间(CI)为0.319~0.755], P=0.0011。支持性分析表明,索凡替尼能够显著延长盲法独立审查委员会(BIIRC) 评估的 PFS, 索凡替尼和安慰剂组分别为 13.9 个月和 4.6 个月, 风险比(HR) 为 0.339 [95%可信区间 (CI) 为 0.209~0.549], P<0.0001。此外, 索凡替尼在 ORR (19.2% vs. 1.9%)、DCR(80.8% vs. 66.0%)等次要研究终点方面也优于安慰剂 组。索凡替尼的安全性和耐受性良好,治疗相关不良事件与既往早期临床研究一 致,最常见的不良反应为蛋白尿、高血压、腹泻等。

索凡替尼是迄今为止, pNET 和 ep-NET 治疗的靶向药物中 ORR 最高(19.2% 和 10%)的药物,在 NET 治疗中显示出良好的疗效与安全性。

# 2. 研究目的和终点

#### 2.1 研究目的

•初步评价索凡替尼联合卡瑞利珠单抗及 mFOLFOX6 方案二线治疗晚期胰腺癌 是否有生存获益,为晚期胰腺癌二线及后线治疗探讨可行性策略。

#### 2.2 研究终点

#### 主要研究终点:

客观缓解率 (ORR)

#### 次要研究终点:

总生存期(OS)、客观缓解率(ORR)、疾病控制率(DCR)、缓解持续时间(DOR)、 总生存期(OS)、生活质量评分、安全性

#### 3. 研究设计

#### 3.1 总体设计

本研究为一项单臂、多中心临床研究,分为二线治疗和二线维持治疗阶段。 拟初步评价索凡替尼联合卡瑞利珠单抗及 mFOLFOX6 方案二线治疗晚期胰腺癌 是否有生存获益,为晚期胰腺癌二线及后线治疗探讨可行性策略。



#### 4. 受试者的选择和退出

#### 4.1 入选标准

患者必须符合以下所有条件才能入组本研究:

- 1. 对本研究已充分了解并自愿签署知情同意书;
- 2. 年龄≥18 岁且≤75 岁, 男女不限;
- 3. 经组织或细胞学确诊的转移性胰腺癌患者;
- 4. 既往接受过一线吉西他滨为基础的化疗失败的患者或前期进行新辅助/辅助治疗期间或治疗结束后 6 个月以内出现疾病进展/复发,,则认为一线全身化疗失败;新辅助/辅助治疗方案同样为吉西他滨为基础的化疗。;
- 5. 患者需至少具有一个可测量病灶(RECIST 1.1);
- 6. ECOG PS 0-1 分;
- 7. 预期生存≥12 周;
- 8. 有潜在生育能力的受试者,需要在研究治疗期间和研究治疗结束后 180 天内 采用至少一种经医学认可的避孕措施(如宫内节育器,避孕药或避孕套);且 在首次用药前血清 HCG 检查必须为阴性;而且必须为非哺乳期。

#### 4.2 排除标准

患者若符合以下任何一项标准,将不得进入本研究:

- 1.28 天内参加过其他抗肿瘤药物临床试验;;
- 2. 既往接受过任何抗 PD-1 抗体、抗 PD-L1 抗体、抗 PD-L2 抗体或抗细胞毒 T 淋巴细胞相关抗原-4(CTLA-4)抗体或作用于 T 细胞协同刺激或检查点通路的任何其它抗体(如 OX40、CD137 等)治疗;
- 3. 既往接受过抗血管内皮生长因子/血管内皮生长因子受体(VEGF/VEGFR)靶向药物治疗:
- 4. 已知对研究中的任何药物存在过敏者;
- 5. 伴有症状或症状控制时间<2 个月的脑转移;
- 6.5年內受试者既往或同时患有其它恶性肿瘤(已治愈的皮肤基底细胞癌和宫颈原位癌除外);
- 7. 骨髓造血功能不足(14天内未输血状态下)::
  - a) 绝对中性粒细胞计数 (ANC) <1.5×10 <sup>9</sup>/L;
  - b) 血小板<100×10 <sup>9</sup>/L;
  - c) 血红蛋白<8g/dL。

#### 8. 肝脏异常;

- a) 无肝转移时,ALT、AST 或 ALP>2.5×正常值参考范围上限(ULN);肝转移时,ALT、AST 或 ALP>5×ULN;
- b) 血清总胆红素>1.5 \*ULN (Gilber 综合症者>3 \*ULN);
- c) 失代偿期肝硬化(Child-Pugh 肝功能评级为B或C级);
- d) 乙肝表面抗原(HBsAg)阳性且乙型肝炎病毒 DNA 拷贝数≥2000IU/mL (HBsAg 阳性且乙型肝炎病毒 DNA 拷贝数<2000IU/mL 者需至少接受 2 周 抗 HBV 治疗才能首次给药);
- e) 丙型肝炎病毒 (HCV) 抗体阳性且 HCVRNA 检测阳性。

#### 9. 肾脏异常:

- a) 血清肌酐>1.5×ULN 或 Cockcroft-Gault 肾小球滤过公式估算的肌酐清除率<60mL/分钟:
- b) 尿常规提示尿蛋白≥++, 且证实 24 小时尿蛋白定量>1.0g;
- c) 肾功能衰竭需要血液透析或腹膜透析;
- d) 既往肾病综合征病史。

#### 10. 出血风险:

- a) 凝血功能异常: 部分活化凝血酶原时间(APTT)或凝血酶时间(TT)>1.5×ULN, 或国际标准化比值(INR)>1.5(需要抗凝治疗的受试者>2.5):
- b) 患有出血(咯血)、凝血性疾病或正在使用华法林、阿司匹林、低分子 肝素及其他抗血小板凝集药物(阿司匹林≤100mg/d 预防性用药除外);
- c) 活动性胃肠道出血,表现为在过去3个月内有呕血、便血或黑便,根据内窥镜或结肠镜检查没有消退证据;
- d) 在首次给药前 4 周内, 出现任何 CTCAE ≥ 3 级出血或流血事件。

#### 11. 心血管异常:

- a) 首次给药前 12 个月内有下列任何情况的受试者: ≥II 级心肌缺血或心肌梗死、心律失常, ≥III 级心功能不全, 未控制的心绞痛, 冠状动脉/周围动脉旁路移植手术, 有症状的充血性心力衰竭, 脑血管意外或短暂性脑缺血发作等;
- b) 首次给药前 6 个月内有深静脉血栓或肺栓塞;

- c) 多普勒超声评估的左室射血分数(LVEF) <50%;
- d) Fridericia 校正后的 QTc 间期(QTcF)平均值(获得至少连续 3 次心电图检测): 男性≥450ms, 女性≥470ms;
- e) 存在药物未能控制的高血压(至少有 2 次测量结果为收缩压 ≥150mmHg, 舒张压≥100mmHg)。
- 12. 免疫缺陷病史:
  - a) 己知人类免疫缺陷病毒(HIV) 感染;
  - b) 其他获得性、先天性免疫缺陷疾病;
  - c) 准备进行或既往接受过器官移植,或首次用药前 60 天内接受过造血干细胞移植,或具有明显的宿主移植反应;
  - d) 需使用免疫抑制剂、或全身、或可吸收的局部激素治疗以达到免疫抑制目的,并在首次给药前7天内仍需继续使用的患者(糖皮质激素每日剂量<10mg、泼尼松或其他等疗效激素除外)。
- 13. 活动性或未能控制的严重感染;
- 14. 受试者存在不能口服药物的情况:
- 15. 研究者认为受试者存在任何临床或实验室检查异常或其他原因而不适合参加本临床研究。

#### 4.3 脱落标准

所有签署了知情同意书,筛选合格进入研究的受试者,均有权随时退出本研究。

- 1. 对于只签署了知情同意书,筛选合格而没有入组的患者,不作为脱落病例。
- 2. 入组后,只要没有完成一个周期的试验无法进行有效性评价者,均为脱落病例。但是由于以下原因除外:
- (1) 入组后因为疾病进展并且有明确的医学证据的,不视为脱落,但是必须提供影像学证据;
  - (2) 因为受试者怀孕或者毒性不可耐受出组者,也不得视为脱落;
  - (3) 研究者从受试者的最大利益出发判定应终止治疗;
  - (4) 入组后死亡。

对于脱落病例,研究者必须记录脱落原因,尽可能完成有关肿瘤评估项目,并且记录末次访视情况。

# 4.4 受试者终止治疗标准

受试者出现以下的任何一种情况,必须停止治疗,但可继续在研究中接受监测:

- 1. 影像学证据表明肿瘤进展;
- 2. 受试者撤回知情同意,要求退出研究;
- 3. 无法耐受毒性者;
- 4. 受试者依从性不佳;
- 5. 受试者失访;
- 6. 研究者认为有必要退出研究的情况。

# 5. 研究实施

# 5.1 研究药物

表 1. 研究药物

| | 索凡替尼 | 卡瑞利珠单抗 |
|---------------------------------------|----------------|--------------------|
| 生产厂家 | 和记黄埔医药(苏州)有限公司 | 苏州圣迪亚生物医药有限公司 |
| \ | | N / / N |
| 剂型 | 胶囊 | 注射液 |
| 规格 | 50mg | 200mg/ 瓶 |
| 用法 | 口服 | 静脉输注 |
| | | 本品从冰箱取出后应立即复溶 |
| | | 和稀释。稀释后药液在室温条 |
| <br> 储存条件 | 遮光、密封,常温(10- | 件下, 贮存不超过 6 小时(包 |
| 间 行 录 门 | 30℃)保存。 | 含输注时间);在冷藏(2-8 ℃ ) |
| | | 条件下,贮存不超过 24 小 |
| | | 时。 |

#### 5.2 给药剂量和方法

#### 5.2.1 给药剂量

每6周(±7天)评估一次疗效,用药超过24周的患者,每12周(±7天)进行1次疗效评价。疾病控制(CR+PR+SD)且不良反应可以耐受的受试者,可持续用药,直到失去临床获益、毒性不可耐受、疗效评价为进展(PD)或免疫治疗证实的疾病进展(iCPD)、研究者认为不适合继续用药时研究结束(以先出现者计)。

- 索凡替尼:索凡替尼推荐日剂量为 250mg,每日一次,连续给药;
- 卡瑞利珠单抗: 给药剂量固定为 240mg, 在联合用药期间每 14 天给药一次, 维持治疗期间每 21 天给药一次, 用药最多满 2 年后停药;
- 化疗方案(mFOLFOX6, 奥沙利铂+亚叶酸钙+氟脲嘧啶): 奥沙利铂
  85mg/m²d1+CF 400mg/m²d1+5-FU 400mg/m²d1/2400mg/m² 持续静注(civ)46h, 每 14 天给药一次, 共 8-12 个周期, 具体周期数由研究者综合判断。

#### 5.2.2 剂量调整

#### 5.2.2.1 剂量调整的一般原则

- 研究期间可根据研究药物的毒副作用对研究药物进行剂量调整,包括:剂量暂停、剂量下调及剂量终止。
- 同时发生不同严重程度级别的不良反应时,应根据观察到的最高级别进行调整。
- 如研究者认为不良反应仅由于研究治疗的一种药物所致,则不需要对另一种药物进行给药调整。
- 对于研究中认为不可能发展为严重或威胁生命的毒性事件,研究治疗可在同一剂量水平,无需减量。
- 在整个治疗研究期间,当受试者因无法耐受某一种药物的不良反应而永久性停用该药物时,若根据研究者判断受试者仍有可能从单药使用中获益,受试者可接受单药治疗,直至符合方案规定的治疗终止标准的事件发生。

#### 5.2.2.2 索凡替尼剂量调整

不良事件处理原则如下文。

表 2. 索凡替尼的剂量调整

| 索凡替尼 | 推荐剂量 |
|---------|-------------|
| 起始剂量 | 250mg QD 口服 |
| 第一次剂量减少 | 200mg QD 口服 |
| 第二次剂量减少 | 150mg QD 口服 |

#### 表3. 针对血液学毒性的剂量调整

| NCI CTCAE v5.0 毒性级别 | 措施 |
|--------------------------------|---------------|
| 1 级或 2 级 | 无 |
| 3 级或 4 级 b | |
| 预期减量后可处理/可逆 | 暂停 a |
| 3 或 4 级毒性 28 天恢复至≤1 级或基线<br>水平 | 降低一个剂量水平 |
| 3级毒性复发 | 降低一个剂量水平或终止治疗 |
| 4级毒性复发 | 终止治疗 |
| <b>3级或4级</b><br>预期减量后不可处理/不可逆 | 终止治疗 |

- a 暂停给予研究药物直至毒性恢复至≤1 级或基线水平。对于毒性缓解超过 28 天的患者,一般需终止治疗,除非研究者认为患者仍可从临床研究中获益。
- b 白细胞或中性粒细胞降低达 3 级或 4 级并在 28 天内恢复到 1 级或基线水平后,则维持原剂量给药。仅当出现中性粒细胞减少症,包括发生>7 天的复发性/持续性 4 级中性粒细胞减少症,或同时伴有发烧或感染,则降低剂量。

表 4. 索凡替尼对非血液学毒性的剂量调整

| NCI CTCAE v5.0 毒性级别 | <b>措施</b> |
|------------------------|-----------|
| 1级或2级(可耐受) | 无 |
| 2级(不可耐受) d | 暂停° |
| 毒性 28 内天恢复至≤1 级或基线水平复发 | 降低一个剂量水平 |

#### 3级或4级d

预测减量后可处理/可逆

3 级毒性 28 天内恢复至≤1 级

3级毒性复发

降低一个剂量水平或终止治疗

暂停°

降低一个剂量水平

4级毒性复发

终止治疗

3级或4级预期减量后不可处理

终止治疗

c 对于毒性持续超过 28 天且未恢复的患者通常需终止该研究,除非研究者确定患者仍能从该研究中获得临床益处。

d 对于恶心、呕吐或腹泻,需先给予支持性治疗,如仍不可耐受,则暂停给予研究药物直至毒性恢复至≤1级或基线水平。另外,对于研究者认为不可能发展为严重或危及生命的毒性事件的毒副反应且患者可耐受(如高尿酸血症、低磷酸盐血症和脱发)。在积极给予对症处理的前提下,研究治疗可维持在同一剂量水平,无需减量。

#### 5.2.2.2.1 索凡替尼常见不良反应的对症处理指南

#### 高血压

对于研究中出现3级或3级以上高血压或血压升高的患者,随后应增加血压监测频率,每周进行血压监测直到血压恢复正常。

| AE级别及定义 | 剂量调整方案 | 处理意见 |
|------------------|--------|-----------------|
| 1级:高血压前期(收缩 | 维持原有剂量 | 无 |
| 压为120-139 mmHg或舒 | | |
| 张压为80-89 mmHg) | | |
| 2 级: 收缩压为140-159 | 维持原有剂量 | 治疗目标: 使血压控制在 |
| mmHg或舒张压为90-99 | | 140/90 mmHg之内*。 |
| mmHg; 或者舒张压症状 | | 若患者基线已接受降压治 |
| 性增加>20 mmHg 或者既 | | 疗,则增加降压给药剂量 |
| 往正常范围,增 | | 或调整降压药物; 若患者 |

| 加>140/90 mmHg; 需要 | | 基线未接受降压治疗,则 |
|-------------------|----------------|-----------------|
| 单药治疗。 | | 使用单一降压疗法。降压 |
| | | 药物的使用或调整,请参 |
| | | 照抗高血压药物的治疗指 |
| | | 南,必要时请心内科医生 |
| | | 会诊 |
| 3 级: 收缩压≥160 mmHg | 降压药物治疗或调整 | 治疗目标: 使血压控制在 |
| 或舒张压为≥100 mmHg; | 降压药物后血压 | 140/90 mmHg之内*。 |
| 或应用一种以上的降压药 | 仍超160/100 mmHg | 开始降压治疗/或增加目前 |
| 物 | 并持续3天以上的, | 的降压药物用量/或增用其 |
| | 暂停索凡替尼治疗; | 他降压药物;降压药物的 |
| | 28天之内能恢复至 | 使用或调整,请参照高血 |
| | 1级或基线水平,降 | 压治疗指南,必要时请心 |
| | 低1 次剂量水平 | 内科医生协助。 |
| 4 级: 致死性结果(如恶 | 终止治疗 | 紧急医学干预 |
| 性高血压、暂时或永久性 | | |
| 神经缺陷及高血压危象) | | |

<sup>\*</sup>对于高风险人群,例如伴有慢性肾脏疾病,伴有糖尿病的患者,或者研究治疗后出现蛋白尿的患者,推荐将血压控制在 130/80 mmHg 的范围内

#### 蛋白尿

如果受试者在治疗期间尿液分析检测发现尿蛋白 2+,请一周内收集 24 小时尿液进行定量检测,根据 24 小时尿液定量检查结果调整索凡替尼剂量。对于蛋白尿≥2+的患者,在随后的 3 个月内应增加尿常规频监测率,即每周进行尿常规检测,若因客观原因,受试者无法至研究中心进行尿液检查,允许在当地二级及二级以上的医院就诊,并及时提供检查报告单(报告单上应有检查项目的正常值范围)。

| AE级别 | 剂量调整方案 | 处理意见 |
|-------------|--------|-------|
| 1级:尿常规检查示尿蛋 | 维持原有剂量 | 按计划随访 |

| 白+; 24小时尿蛋白定量 | | |
|-------------------|----------------|-------------|
| 检测<1.0g | | |
| 2 级: 尿常规检查示尿蛋 | 积极保肾治疗,可维持积 | 积极治疗并监测尿常规 |
| 白++或以上;24小时尿蛋 | 原剂量继续治疗 | (每周1次),必要时 |
| 白定量检测 1.0g - 2.0g | | 请 |
| (不含2.0 g) | | 肾内科医生会诊 |
| 2 级: 尿常规检查示尿蛋 | 首次出现: 暂停用药, 28 | 积极治疗并监测尿常规 |
| 白++或以上; 24小时尿蛋 | 天之内能恢复至≤1级,维 | (每周1次),必要时 |
| 白定量检测2.0 - 3.5g(不 | 持原剂量给药,如果恢复 | 请肾内科医生会诊。 |
| 含3.5g) | 时间超过28天若研究者判 | |
| | 断仍有获益,与资助方商 | |
| | 定后,需降低一个剂量给 | |
| | 药 | |
| | 再次出现: 暂停用药, 28 | |
| | 天之内能恢复至≤1级,降 | |
| | 低一个剂量给药; | |
| | 如果恢复时间超过28天, | |
| | 与资助方商定(降低一个 | |
| | 剂量给药或终止治疗)。 | |
| 3 级: 24小时尿蛋白定量 | 暂停用药,28天之内能 | 积极治疗并监测尿常规 |
| 检测 ≥3.5g | 恢复至1级,降低一个剂量 | (每周1-2次),必要 |
| | 水平重新给药。如果恢复 | 时 |
| | 时间超过28天,与申办方 | 请肾内科医生会诊。 |
| | 商定(降低一个剂量给药 | |
| | 或终止治疗)。 | |

# 肝功能损伤的剂量调整方案

肝功能异常(包括 ALT 升高,或 AST 升高或总胆红素升高等具有临床意义

的指标异常)的剂量调整方案\*:

| AE级别 | 剂量调整方案 | 处理意见 |
|---------------------|---------------|-------------|
| 1级: ALT>ULN-3ULN或 | 维持原有剂量 | 按计划随访 |
| AST>ULN-3ULN | | |
| 2级: ALT>3.0-5.0ULN或 | 维持原有剂量,经保肝治 | 积极保肝治疗并监测肝 |
| AST>3.0-5.0ULN | 疗,观察1周,若转氨酶 | 功能(每周1-2次)。 |
| | 稳定或下降,则继续原剂 | |
| | 量治疗; 若转氨酶明显继 | |
| | 续升高,则暂停研究药 | |
| | 物,28天之内恢复至≤1级 | |
| | 或基线水平,维持原剂量 | |
| | 给药。 | |
| 3级: ALT>5.0-20.0ULN | 首次出现:暂停用药,28 | 积极保肝治疗并监测肝 |
| 或AST>5.0-20.0ULN | 天之内能恢复至<1级或基 | 功能(每周2次),必要 |
| | 线水平,需降低一个剂量 | 时请医生会诊; |
| | 给药;如果恢复时间超过 | |
| | 28天,一般需终止治疗。 | |
| 4级: ALT>20.0ULN或 | 终止治疗 | 紧急医学干预 |
| AST>20.0ULN | | |

\*"需要立即停药,并立即向申办方报告的肝功能异常包括:1.基线时肝功能异常(ALT、AST和胆红素均在正常范围内)的患者,在同一次采集的血样中,测得AST和/或ALT升高 >3倍ULN,合并血清总胆红素升高>2倍ULN。2.基线时转氨酶已升高的患者,在同一次 采集的血样中,测得AST和/或ALT升高>基线值的2倍,合并血清总胆红素升高>2倍 ULN。

#### 任何部位出血的剂量调整方案

| AE级别 | 剂量调整方案 | 处理意见 |
|------|--------|------|
|------|--------|------|

| 1级 | 原有剂量水平 | 按计划随访 |
|------|-----------------|--------|
| 2级 | 暂停用药;28天之内能恢复至1 | 积极处理 |
| | 级或以下的,降低一次剂量水平 | |
| ≥3 级 | 终止治疗 | 紧急医学干预 |

# 5.2.2.3 卡瑞利珠单抗剂量调整

根据个体患者的安全性和耐受性,可能需要暂停给药或永久停药。不建议增加或减少剂量。有关暂停给药和永久停药的指南,请见表 5 所述。有关免疫相关性不良反应管理的详细指南,请参见【注意事项】。。

表 5. 推荐的卡瑞利珠单抗针治疗调整方案

| | 严重程度: | 治疗调整方案 |
|---|---|---|
| 反应性毛细血管增生症* | 3 级 | 暂停用药,至不良反应恢<br>复至 0-1 级 |
| | 4 级 | 永久停药 |
| 免疫相关不良反应 | | |
| 肺炎 | 2 级 | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| | 3级或4级或复发性2级 | 永久停药 |
| 腹泻及结肠炎 | 2 级或 3 级 | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| | 4 级 | 永久停药 |
| 肝炎<br>(适用于非肝细胞癌患<br>者) | 2 级,天门冬氨酸氨基转移酶<br>(AST)、丙氨酸氨基转氨酶<br>(ALT)在 3-5 倍正常值上限<br>(ULN)或总胆红素(TBIL)<br>在 1.5-3 倍 ULN | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| | 3 级或 4 级,AST、ALT>5 倍<br>ULN,或总胆红素>3 倍 ULN | 永久停药 |
| 肝炎 | AST 或 ALT: 3-5 倍 ULN,若基线状态在正常范围内 | 暂停给药,直至不良反应<br>恢复至 0-1 级或者至基线 |

| | 严重程度: | 治疗调整方案 |
|---|---|---|
| (适用于肝细胞癌患者) | AST 或 ALT: 5-10 倍 ULN,<br>若基线状态 AST 或 ALT 在 1-<br>3 倍 ULN | 状态后恢复给药 |
| | AST 或 ALT: 8-10 倍 ULN,<br>若基线状态在 3-5 倍 ULN | |
| | 总胆红素: 1.5-3 倍 ULN | |
| | AST 或 ALT: >5 倍 ULN,若基线状态在正常范围内 | |
| | AST 或 ALT: >10 倍 ULN,若基线状态>ULN | 永久停药 |
| | 总胆红素>3 倍 ULN | |
| 肾炎 | 2级或3级血肌酐升高 | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| | 4级血肌酐升高 | 永久停药 |
| | 症状性 2 级或 3 级甲状腺功能减退、2 级或 3 级甲状腺功能亢进、2 级或 3 级垂体炎、2 级肾上腺功能不全 | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| | 3 级高血糖症或糖尿病 | |
| 内分泌疾病 | 4级甲状腺功能减退<br>4级甲状腺功能亢进 | |
| | 4 级垂体炎 | 永久停药 |
| | 3级或4级肾上腺功能不全 | |
| | 4级高血糖症或糖尿病 | |
| | 3 级 | 暂停给药,直至不良反应<br>恢复至 0-1 级 |
| 皮肤不良反应 | 4级,史蒂文斯—约翰逊综合征<br>(SJS)或中毒性表皮坏死松解<br>症(TEN) | 永久停药 |
| 血小板减少症 | 3 级 | 暂停给药,直至不良反应 |

| | 严重程度‡ | 治疗调整方案 |
|---|---|---|
| | | 恢复至 0-1 级 |
| | 4级 | 永久停药 |
| | 3级或4级血淀粉酶升高或脂肪酶升高 | |
| | 2级或3级胰腺炎 | 暂停给药,直至不良反应 |
| | 2级心肌炎** | 恢复至 0-1 级 |
| 其他免疫相关不良反应 | 2 级或 3 级首次发生的其他免疫相关性不良反应 | |
| 兴也九汉相八 <b>个</b> (次)点 | 4 级胰腺炎或任何级别的复发性胰腺炎 | |
| | 3级或4级心肌炎 | 永久停药 |
| | 3级或4级脑炎 | <b>小八</b> 厅约 |
| | 4 级首次发生的其他免疫相关性不良反应 | |
| | 复发性3级或4级(内分泌疾病除外) | |
| 复发或持续的不良反应 | 末次给药后 12 周内 2 级或 3<br>级不良反应未改善到 0-1 级<br>(内分泌疾病除外) | 永久停药 |
| | 末次给药后 12 周内皮质类固醇未能降至≤10 mg/天强的松等效剂量 | |
| 输液反应 | 2 级 | 降低滴速或暂停给药,当<br>症状缓解后可考虑恢复用<br>药并密切观察 |
| | 3 级或 4 级 | 永久停药 |

参考卡瑞利珠单抗注射液说明书。

‡不良反应严重程度依据美国国立癌症研究所的不良事件通用术语评估标准第 4.03 版 (NCI-CTCAE v4.03)。

\*反应性毛细血管增生症分级依据《CSCO 免疫检查点抑制剂相关的毒性管理指南 2019》。

\*\*心肌炎经治疗改善到 0-1 级后重新开始本品治疗的安全性尚不明确。

注:不良反应严重程度依据美国国立癌症研究所的不良事件通用术语评估标准第 4.03 版 (NCI-CTCAE v5.0)。

#### 5.2.2.4 化疗剂量调整

对于化疗引起的不良反应,由研究者决定剂量调整方案。

#### 5.2.2.5 联合用药调整

对于联合用药共有的或临床无法判定由哪个单药引起的不良反应,由研究者判断相关性,决定减量或停用哪个药物。

# 6. 研究程序

#### 6.1 筛选评估(-28~0天)

**所有筛选评估步骤前应获得受试者签字的知情同意书。**以下筛选评估的程序 应筛选期(第-28~0 天)内完成。这些评估的计划和类型详情如下:

- 核对入选/排除标准:
- 记录人口学数据:
- 既往病史、既往用药和合并用药:
- 不良事件记录:
- 身高、体重、生命体征(体温,脉搏,呼吸频率,血压);
- ECOG评分;
- 体格检查:一般情况,头面部,皮肤,淋巴结,眼(巩膜、瞳孔),耳部,鼻部,咽喉部,口腔、呼吸系统,心血管系统,腹部(包含肝脾),生殖-泌尿系统,肌肉骨骼,神经系统,精神状况;(注:试验期间须进行全面的体格检查,只需记录异常情况,如与筛选期相比无变化,则不需重复记录);
- 实验室检查:血常规,血生化,尿常规,大便常规,凝血功能,甲状腺功能, 血HCG检测(有潜在生育能力的受试者); HBV, HCV, HIV检查;
- 十二导联心电图:
- 心脏超声检查;
• 影像学评估:胸部+腹部+盆腔CT增强扫描。如存在造影剂过敏等其他原因不能耐受增强扫描受试者,应采用MRI检查;

### 6.2 治疗期

受试者筛选成功后进入治疗期。受试者必须在特定的时间点进行相关评价和流程安排(参见研究流程表)。每个治疗周期为 2 周/3 周(治疗阶段为 2 周,维持阶段为 3 周),入组受试者将接受索凡替尼联合卡瑞利珠单抗和 mFOLFOX6 化疗方案治疗。可持续给药至每次来院需收发研究药物及受试者日志卡,统计实际服药量,评价受试者的服药依从性。

- 不良事件及合并用药;
- 生命体征(体温,脉搏,呼吸频率,血压)、体重:第一周期 D1,之后每 2 周或 3 周检查一次;
- ECOG 评分:第一周期 D1,之后每 2 周/3 周检查一次;
- 体格检查: 第一周期 D1, 之后每 2 周/3 周进行症状为导向的体格检查:
- 给予研究药物:索凡替尼每日口服一次,需填写用药日志卡;
- 血常规, 血生化, 尿常规、大便常规: 每周期 D1±7 天内进行;
- 凝血功能、甲状腺功能:每两周期 D1±7 天内进行:
- 十二导联心电图:每周期 D1±7 天内进行;心电图显著异常者,研究者根据 受试者情况加查心脏超声;
- 影像学评估:每6周/12周±7天进行一次(治疗阶段每6周(±7天)接受一次肿瘤影像学评估,用药超过24周的患者,每12周(±7天)进行1次疗效评价。
- 研究期间的所有血标本或组织标本的检测地点为中山大学附属肿瘤医院,同时,受试者就诊检查所产生的医疗废弃物按照中心常规医疗废物处置管理制度执行清理。受试者的生物标本将仅用于科研探索,研究者将确保受试者的样本信息安全。

### 6.3 治疗结束/退出研究评估

如受试者满足任何停药标准,受试者应终止研究治疗。研究结束时应进行相关检查,详见流程图。

### 6.4 随访期

### 6.4.1 安全性随访

所有受试者末次用药后 30 天,均需到研究中心进行安全性随访。具体访视 内容见流程图。

### 6.4.2 生存随访

受试者完成停止给药后 30 天的访视,则进入生存期随访。因除疾病进展以外的原因停止用药的受试者,按照既定时间继续进行影像学评估,直至进展、开始新的抗肿瘤治疗、撤回知情同意、失访、死亡或研究结束(以先发生者为准)。应每 3 个月(±7 天)实施一次生存评估。可通过电话联系受试者、受试者家人,收集生存数据,直至受试者死亡、撤回知情同意、失访或研究结束(以先发生者为准)。

# 7. 研究评价和程序

## 7.1 基线评估

描述所有人口统计学和基线数据。描述统计表中连续变量数据包括: 受试者例数、均值、中间值、标准差以及范围(极小值-极大值)。频率统计表中分类变量数据包括: 受试者例数、比例。

# 7.2 安全性评估

进行以下评估以衡量其安全性和耐受性:

临床实验室检查(采集血样、尿样用于临床实验室参数检查)、ECOG 体力 状态评分、体格检查(包括生命体征测量)、ECG 以及治疗相关不良事件的 发生率和严重程度。

## 7.3 有效性评估

筛选时的首次肿瘤影像学检查必须在入组前 28 天内进行。研究者应确认受试者至少具有一个符合 RECIST (1.1 版)标准的可测量病灶。RECIST (1.1 版)评估方法见附录 1。

整个研究期间,应尽量按照方案规定的影像学评估计划时间点进行评估。自用药开始,治疗阶段每6周(±7天)接受一次肿瘤影像学评估,用药超过24周的患者,每12周(±7天)进行1次疗效评价;一线维持治疗阶段,若维持治疗为索凡替尼联合卡瑞利珠单抗,每8周(±7天)接受一次肿瘤影像学评估。直至疾病进展、撤销知情同意或研究结束。如怀疑新发病灶可适时检查;首次评价PR/CR受试者须在至少4周(±7天)后进行疗效确认。

对于非影像学证据进展的受试者(不可耐受、其他情况),每3个月进行一次肿瘤评估直到疾病进展、死亡或开始其他抗肿瘤治疗。

最佳总体疗效是指从用药开始到按照 RECIST (1.1 版)标准客观记录进展的日期或到开始用后续抗肿瘤治疗的日期(以先发生者为准)这段时间内记录的最佳疗效。

# 8. 不良事件报告

### 8.1 不良事件定义(AE)

不良事件是病人或临床试验的受试者接受一种药品后出现的不良医学状况或已有医学状况恶化,但不一定与治疗有因果关系。按照 GCP 的要求,不管是否与试验用药有因果关系,研究者均应在原始记录中记录所有不良事件,并转抄至病例报告表中。术语"不良事件"包括了严重不良事件和非严重不良事件。

# 8.2 不良事件的记录

1)不良事件描述; 2)发生时间; 3)终止时间; 4)发作程度及频度; 5)是否需要治疗,如需要,请记录所给予的治疗; 6)研究者判断不良事件是否与应用试验药品有关。

发现不良事件时,观察医师可根据病情决定是否终止观察,不良事件应追踪至解决。有关不良事件的医学文件均应记录在原始文件中,包括实验室检查的通知单(如: X 线检查、心电图等)和检查结果报告单。如受试者因试验结束或受试者出院等而无法继续接受研究者的治疗,研究者应将受试者的病例摘要(包括治疗安排和不良事件是否需要继续随访的说明等)交给负责继续治疗他们的医生。这些信息也要求记录在原始文件中。

## 8.3 不良事件的程度

不良反应按抗癌药物常见毒副反应分级标准(NCICTCAE 5.0 版分级标准)。如 NCI 毒性分级标准未列出的不良事件,可根据以下标准判断:

- 1级:轻度,无临床症状或有轻微临床症状;仅有临床或实验室检查异常;不需治疗。
- 2级:中度,需要微量的、局部的或非侵害性的治疗,与年龄相符的使用工具的 日常生活活动(ADL)受限,如做饭、扫地、数钱等:
- 3级:病情严重或有医学上严重的症状但暂时不危及生命;导致住院或住院时间延长;日常生活自理受限,如洗澡、穿衣、吃饭、上厕所、吃药等。
- 4级: 危及生命, 需紧急治疗。
- 5级: 因不良事件致死。

## 8.4 不良事件与药物的相关性评价

# 不良事件判断表

| 判断结果 - | | 判 | 断 指 | 标 * | |
|--------|---|---|-----|-----|---|
| | 1 | 2 | 3 | 4 | 5 |
| 肯定有关 | + | + | | + | + |

| 很可能有关 | + | + | | + | ? |
|-------|---|---|---|---|---|
| 可能有关 | + | + | ± | ± | ? |
| 可能无关 | + | _ | ± | ± | ? |
| 肯定无关 | _ | _ | ± | _ | |

注: +表示肯定, --表示否定, ±表示难以肯定或否定, ?表示情况不明

不良反应判断①肯定有关:同时符合上述第 1、2、4、5 条标准;②很可能有关:同时符合上述第 1、2、4 条标准;③可能有关:同时符合上述第 1、2 条标准;④可能无关:符合上述第 1 条标准;⑤肯定无关:上述 5 条标准中,一条也不符合。

- ①肯定有关、很可能有关、可能有关三级可判断为不良反应。② 实验室检查项目超过正常值的 20%判为异常。
- \*不良事件判断指标(包括症状、体征、试验指标)
- 1)不良事件出现的时间与用药时间吻合; 2)不良事件与该药的已知不良反应有关; 3)不良事件不能用其它原因解释; 4)不良事件在停药后消失; 5)不良事件在给药后再现。

### 8.5 严重不良事件(SAE)

严重不良事件(SAE)指受试者接受试验用药品后出现死亡、危及生命、永久或者严重的残疾或者功能丧失、受试者需要住院治疗或者延长住院时间,以及先天性异常或者出生缺陷等不良医学事件。

- 应快速报告的其他事件:
- 1、妊娠/哺乳期的药物接触。原则上,妊娠和哺乳期属于入选排除标准。如研究期间女性受试者或男性受试者的女性伴侣发生妊娠,那么患者应立刻退出研究,并应立即告知研究者,并且对患者在整个妊娠期及产后进行随访。即使母子均完全正常没有任何不良事件,也应对其后果进行记录。即使妊娠不属于 SAE,也应使用妊娠报告表并在研究者获知的 24 小时内报告。
- 2、方案规定的特殊不良事件。以下事件为方案规定的特殊事件,无论是否为 SAE,均须在研究者获悉的 24 小时内报告。

肝功能异常:在受试者/患者同一次采集的血样中,测得转氨酶[丙氨酸氨基转移酶(ALT)和/或天门冬氨酸氨基转移酶(AST)]≥3倍正常值上限(ULN)合并总胆红素≥2倍ULN 出血:CTCAE3级或以上

• 不应作为 SAEs 来处理的事件:

疾病进展一般不判断为 SAE (但如果疾病进展的症状和体征满足 SAE 的标准,则可以报告为 SAE)。

死亡本身是一种后果,不被视为 SAE (应将死亡的主要原因,即导致死亡的主要 AE 记录和报告为 SAE,将"死亡"报告为相应 AE 的后果;如果死亡没有确切的原因可以报告,则可将死亡本身报为 SAE)。

受试者开始用药至末次用药 30 天内开始新的抗肿瘤治疗前出现死亡应作为 SAE 上报,如果是因疾病进展导致的死亡,则将不作为 SAE 报告。此后,仅报告与研究药物相关的死亡。

在本研究中由于疾病的严重性,某些被确定为 SAEs 的情况可能需从即刻报告中排除:

A.事先计划的的住院和手术治疗

B.可选择的住院治疗,目的为简化治疗或研究措施,而非不良事件本身导致的住院

# 9. 统计学分析

# 9.1 样本量确定

查阅文献知历史对照 ORR: 胰腺癌二线治疗 ORR 为 6%-15%左右,参考多个二线治疗研究结果并结合临床时间,选择 ORR 为 10%作为历史数据参考,假设卡瑞利珠单抗联合化疗和靶向的 ORR 为 25%。单侧检验,取I类错误 0.05,基于 0.80 的功效,使用 PASS 软件计算样本量。考虑脱落率 10%,样本量需放大至 33/0.9=36.67,向上取整取 37。

### 9.2 统计方法

### 统计分析集:

意向性分析集(Intention-to-treat Analysis Set, ITT): 按照意向性分析(ITT)原则,包含所有入组的患者。

PPS 集(Per-Protocol Set): 包含 ITT 集中未发生影响疗效评估的重大方案偏离的患者。对缺失数据不进行任何填补(imputation)。对药物的疗效同时对 ITT 和 PPS 进行统计分析。

SS 集(Safety Set): 安全性分析数据集。至少接受一次研究药物治疗且至少有一次安全性评估的受试者。该数据集用于安全性分析。

### 9.2.1 有效性分析

有效性分析将基于 ITT 及 PPS 集:

• 客观有效率(ORR):根据 RECIST(1.1 版)标准,发生完全缓解(CR)或部分缓解(PR)的受试者在分析人群中所占的比例(公式如下)。提供 ORR的 95%CI。

$$ORR = \frac{CR + PR$$
的受试者例数 \* 100% 总受试者数

• 无进展生存期(PFS): 定义为受试者从首次用药日期开始,至第一次记录肿瘤进展(按照 RECIST 1.1 标准评定,无论是否继续治疗)的日期或因任何原因死亡的日期,以先出现的为准。

在确定 PFS 时,在无确凿的疾病进展证据(根据 RECIST 1.1)的情况下出现的临床恶化不属于进展。对于以前没有报告进展的死亡受试者,将其视为在死亡日期发生了进展。既没有发生疾病进展也没有死亡的受试者将会在其最后一次可评价的肿瘤评价日期被删失。研究期间没有任何肿瘤评价而且也没有死亡的受试者将会在首次用药日期被删失。由于疾病进展以外的原因而中止研究(无后续影像学检查)的受试者,将以中止研究的时间作为数据删失。之前没有报告疾病进展却开始了后续抗肿瘤治疗的受试者,将会在开始用后续抗肿瘤治疗之前最后一次可评价的肿瘤评价日期、或者开始后续抗肿瘤治疗时被删失。当受试者不是以中止研究的时间或开始接受后续抗肿瘤治疗的时间作为数据删失时,预先计划

的灵敏度统计学分析将仅根据出现影像学证实的进展的事件时间来进一步确认 PFS。新发其他肿瘤不视为疾病进展事件,并且也不作为数据删失。

将采用 Kaplan-Meier 方法分析 PFS,及其 95%CI,并绘制生存曲线图。

•疾病控制率(DCR):根据 RECIST (1.1 版)标准,发生完全缓解(CR)或部分缓解(PR)或疾病稳定(SD)的受试者在分析人群中所占的比例(公式如下)。提供 DCR 的 95%CI。

$$DCR = \frac{CR + PR + SD$$
的受试者例数  $*100\%$  总受试者数

- 持续缓解时间 (DOR): 定义为第一次测量符合 CR 或 PR 的标准 (首次记录未准) 直到客观记录的疾病复发日期或进展日期 (治疗开始后的记录到的最小测量病灶为疾病进展的参照)。
- 总生存期 (OS): 定义为从首次用药日期到因各种原因导致受试者死亡之间的时间。末次随访时仍存活的受试者,其 OS 以末次随访时间计为数据删失。失访的受试者,其 OS 以失访前末次证实存活时间计为数据删失。数据删失的 OS 定义为从首次用药到删失的时间。

将采用 Kaplan-Meier 方法分析 OS,中位 OS 及其 95%CI,并绘制生存曲线图。

## 9.3.2 安全性分析

安全性分析将基于安全性人群的数据。

汇总试验期间发生的不良事件,并按 CTCAEv5.0 分级。此外,不良反应、严重不良事件、严重不良反应、CTCAE v5.0 3 级以上的不良事件、3 级以上的不良反应、导致研究药物暂停、减量、终止的不良事件、任何原因的死亡、特别关注的不良事件将相应地进行汇总。多次发生的相同事件,将按最高严重程度记为1 起事件。按报告至少发生1 件不良事件的受试者比例。将汇总特定实验室检查结果、生命体征、体格检查以及12 导联 ECG 检查值和其相对基线的变化。在适用的情况下,基线检查值与基线后各时间点检查值用交叉表形式呈现。

# 10.数据收集和管理

### 10.1 病例报告表(CRF)

病例报告表(CRF)是临床试验中临床资料的记录方式,主要的目的是以完整、准确、清晰、及时的方式获得研究方案必需的资料。病历报告表中的数据应当与原始文件一致。

病历报告表的填写必须完整、清晰(使用黑色或蓝色原珠笔,符合法定文件要求)。为保证受试者的隐私权,CRF上的受试者姓名需使用代码。所有修订和改正必须有研究者进行和确认,注明修订/改正的日期。错处必须清晰地保留,不能用改正的资料覆盖(例如使用修正液)。研究者必须标明他/她修订重要资料的原因。病历中丢失的资料/附注,在病历报告表中的空格输入应以划线取消来代替,以避免不必要的后续调查。

病历报告表是法规文件, 必须适合提交给医院当局。

### 10.2 数据管理

遵照 ICH/GCP 指南,研究者/机构将维护从每名受试者采集数据的 CRF 和所有源文档、临床研究实施重要文件中规定的所有研究文档,与适用法规要求规定的所有研究文档。研究者/机构将采取措施防止意外或过早销毁这些文档。重要的文档必须加以保留,直至研究药物临床研究正式中止后至少过去 10 年为止。

# 11.伦理道德

# 11.1 研究者的责任

研究者应负责确保临床研究按研究方案执行,伦理道德原则依据赫尔辛基宣言(赫尔辛基的世界医学协会宣言,当前修订版)和药物临床试验管理规范(GCP),并依据中国国情适当进行调整。以上文件必须阐明在受试者的知情同意书上,这是入选临床研究基本的先决条件。

## 11.2 伦理委员会

研究开始前,应该将研究方案以及相关文件(例如受试者信息、知情同意书、研究者手册等)一起交给伦理委员会,并得到他们的同意。伦理委员会同意/批准的研究文件应存档。研究只有在得到书面同意后才能进行。

研究方案的任何修订都应该交付伦理委员会,并根据国际和/或当地要求将严重不良事件报告给 IRB。

## 11.3 受试者信息

签署书面知情同意书是受试者入选必须的前提条件。在签署之前,研究者必 须为受试者提供充足的信息。如果符合医院条规,可以通过被研究者指定执行人 员给受试者提供信息给。除了书面信息以外,研究者或执行人员应口头告知受试者。注意选择措辞,以便受试者能充分、容易地理解。

无论何时,只要发现有重要的新信息且涉及到受试者的知情同意书,受试者信息表应作修改。

# 11.4 知情同意书

在进行所有与研究相关的行为之前,必须有受试者愿意参加临床研究的书面同意书。知情同意书需受试者和研究者/研究者指定的执行人员亲自签署,标明签署日期。

研究者应在 CRF 中再次确认是否签署同意书。已经签署且标明日期的知情同意书应存放在研究者处,必须由研究者安全存档,以便任何时候监督、审核、检查。知情同意书副本原件应在进行研究前提供给受试者。

如果受试者或法律上承认的代表不能阅读知情同意书,那么应该有一名可靠、独立的见证人出席讨论知情同意书的全过程。见证人的选择必须保证受试者保密性的权利。可靠、独立的见证人应该是独立的个体,而不是附属于研究机构或参加研究的人员。家庭成员或熟人是独立见证人的合适选择。如果可能,在受试者或受试者或法律上承认的代表口头同意并签署知情同意书后,见证人应当在知情同意书上亲自签名并标注日期,以证明信息是准确的,因为只有受试者或法律上

承认的代表充分理解知情同意书的内容,才是真正的知情同意书。

# 12. 参考文献列表

- 1. GLOBOCAN 2020
- 2. Zeng H, Chen W, Zheng R, et al. Changing cancer survival in China during 2003-15: a pooled analysis of 17 population-based cancer registries. Lancet Glob Health. 2018 May;6(5):e555-e567.
- 3. Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21.
- 4. Von Hoff DD, Ervin T, Arena FP, et al. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703.
- 5. Conroy T, Desseigne F, Ychou M, et al. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25.
- 6. Chiorean EG, Cheung WY, Giordano G, et al. Real-world comparative effectiveness of nab-paclitaxel plus gemcitabine versus FOLFIRINOX in advanced pancreatic cancer: a systematic review. Ther Adv Med Oncol. 2019 May 19;11:1758835919850367
- 7. Kang J, Hwang I, Yoo C, et al. Nab-paclitaxel plus gemcitabine versus FOLFIRINOX as the first-line chemotherapy for patients with metastatic pancreatic cancer: retrospective analysis. Invest New Drugs. 2018 Aug;36(4):732-741.
- 8. Portal A, Pernot S, Tougeron D, et al. Nab-paclitaxel plus gemcitabine for metastatic pancreatic adenocarcinoma after Folfirinox failure: an AGEO prospective multicentre cohort. Br J Cancer. 2015 Sep 29;113(7):989-95.
- 9. WANG-GILLAM A, LI CP, BODOKY G, et al.Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial.Lancet, 2016, 387 (10018): 545-557.
- 10. Yung-Jue Bang, Chung-Pin Li, Kyung-Hun Lee, et al.Liposomal Irinotecan in Metastatic Pancreatic Adenocarcinoma in Asian Patients: Subgroup Analysis of the

- NAPOLI-1 Study. Cancer Sci, 2020, 111 (2): 513-527.
- 11. Oettle H, Riess H, Stieler JM, et al. Second-line oxaliplatin, folinic acid, and fluorouracil versus folinic acid and fluorouracil alone for gemcitabine-refractory pancreatic cancer: outcomes from the CONKO-003 trial. J Clin Oncol. 2014 Aug 10;32(23):2423-9.
- 12. Yoo C, Hwang JY, et al. A randomised phase II study of modified FOLFIRI.3 vs modified FOLFOX as second-line therapy in patients with gemcitabine-refractory advanced pancreatic cancer. Br J Cancer. 2009 Nov 17;101(10):1658-63.
- 13. Hecht JR, Lonardi S, Bendell J, et al. Randomized Phase III Study of FOLFOX Alone or With Pegilodecakin as Second-Line Therapy in Patients With Metastatic Pancreatic Cancer That Progressed After Gemcitabine (SEQUOIA). J Clin Oncol. 2021 Apr 1;39(10):1108-1118.
- 14. Xu J , Shen L , Bai C , et al. Surufatinib in advanced pancreatic neuroendocrine tumours (SANET-p): a randomised, double-blind, placebo-controlled, phase 3 study[J]. The Lancet Oncology, 2020, 21(11): 1489-1499.
- 15. Xu J , Shen L , Zhou Z , et al. Surufatinib in advanced extrapancreatic neuroendocrine tumours (SANET-ep): a randomised, double-blind, placebo-controlled, phase 3 study[J]. The Lancet Oncology, 2020, 21(11):1500-1512.
- 16. Momeny M, Alishahi Z, Eyvani H, et al. Anti-tumor activity of cediranib, a pan-vascular endothelial growth factor receptor inhibitor, in pancreatic ductal adenocarcinoma cells. Cell Oncol (Dordr). 2020 Feb;43(1):81-93.
- 17. Candido JB, Morton JP, Bailey P, et al. CSF1R+ Macrophages Sustain Pancreatic Tumor Growth through T Cell Suppression and Maintenance of Key Gene Programs that Define the Squamous Subtype. Cell Rep. 2018 May 1;23(5):1448-1460.

## 13. 附件一: 实体瘤疗效评价标准(RECIST 1.1 版)

### 1. 肿瘤在基线水平的可测量性

### 1.1 定义

在基线水平上,肿瘤病灶/淋巴结将按以下定义分为可测量和不可测量两种: **1.1.1 可测量病灶** 

肿瘤病灶: 至少有一条可以精确测量的径线(记录为最大径), 其最小长度如下:

- CT 扫描 10 mm (CT 扫描层厚不大于 5mm)
- 临床常规检查仪器 10 mm(肿瘤病灶不能用测径仪器准确测量的应记录为不可测量)
- 胸部 X-射线 20 mm
- 恶性淋巴结: 病理学增大且可测量,单个淋巴结 CT 扫描短径须≥15 mm (CT 扫描 层厚推荐不超过 5mm)。基线和随访中,仅测量和随访短径。

#### 1.1.2 不可测量病灶

所有其他病灶,包括小病灶(最长径<10 mm 或者病理淋巴结短径≥10 mm 至<15 mm) 和无法测量的病灶。无法测量的病灶包括:脑膜疾病、腹水、胸膜或者心包积液、炎性乳腺癌、皮肤/肺的癌性淋巴管炎、影像学不能确诊和随诊的腹部包块,以及囊性病变。

### 1.1.3 关于病灶测量的特殊考虑

骨病灶、囊性病灶和先前接受过局部治疗的病灶需要特别注明: 骨病灶:

- 骨扫描, PET 扫描或者平片不适合于测量骨病灶, 但是可用于确认骨病灶的存在或者消失;
- 溶骨性病灶或者混合性溶骨/成骨病灶有确定的软组织成分,且软组织成分符合上述可测量性定义时,如果这些病灶可用断层影像技术如 CT 或者 MRI 进行评价,那么这些病灶可以作为可测量病灶:
- 成骨病灶属不可测量病灶。

#### 囊性病灶:

- 符合放射影像学单纯囊肿定义标准的病灶, 不应因其为定义上的单纯性囊肿, 而认为是恶性病灶, 既不属于可测量病灶, 也不属于不可测量病灶;
- 若为囊性转移病灶,且符合上述可测量性定义的,可以作为是可测量病灶。但如果在同一病人中存在非囊性病灶,应优先选择非囊性病灶作为靶病灶。 局部治疗过的病灶:
- 位于曾放疗过或经其他局部区域性治疗的部位的病灶,一般作为不可测量病灶,除非该病灶出现明确进展。研究方案应详细描述这些病灶属于可测量病灶的条件。

### 1.2 测量方法说明

#### 1.2.1 病灶测量

临床评价时,所有肿瘤测量都要以公制米制记录。所有关于肿瘤病灶大小的基线评定都 应尽量在接近治疗开始前完成,且必须在治疗开始前的28天内(4周)完成。

#### 1.2.2 评价方法

对病灶基线评估和后续测量应采用同样的技术和方法。除了不能用影像学检查,而仅能 用临床检查来评价的病灶之外,所有病灶必须使用影像学检查进行评价。

临床病灶: 临床病灶只有位于浅表且测量时直径≥10 mm 时才能认为是可测量病灶(如皮肤结节等)对于有皮肤病灶的受试者,建议用含有标尺测量病灶大小的彩色照片作为存档。 当病灶同时使用影像学和临床检查评价时,由于影像学更客观且研究结束时可重复审阅,应 尽可能选用影像学评价。 胸部 X 片: 当肿瘤进展作为重要研究终点时,应优先使用胸部 CT,因为 CT 比 X 线更敏感,尤其对于新发病灶。胸部 X 片检测仅当被测量病灶边界清晰且肺部通气良好时适用。

CT、MRI: CT 是目前用于疗效评价最好的可用可重复的方法。本指导原则对可测量性的定义建立在 CT 扫描层厚≤5 mm 的基础上。如果 CT 层厚大于 5 mm,可测量病灶最小应为层厚的 2 倍。MRI 在部分情况下也可接受(如全身扫描)。

超声:超声不应作为一种测量方法用于测量病灶大小。超声检查因其操作依赖性,在测量结束后不具备可重复性,不能保证不同测量间技术和测量的同一性。如果在试验期间使用超声发现新病灶,应使用CT或者MRI进行确认。如果考虑到CT的放射线暴露,可以使用MRI代替。

内窥镜,腹腔镜检查:不建议使用这些技术用于肿瘤客观评价,但这种方法在取得的活检标本时可以用于确认 CR,也可在研究终点为 CR 后复发或手术切除的试验中,用于确认复发。

肿瘤标志物: 肿瘤标志物不能单独用来评价肿瘤客观缓解。 但如果标志物水平在基线时 超过正常值上限,用于评价完全缓解时必须回到正常水平。因为肿瘤标志物因病而异,在将测量标准写入方案中时需考虑到这个因素。有关 CA-125 缓解(复发性卵巢癌)及 PSA (复发性前列腺癌)缓解的特定标准已经发表。 且国际妇科癌症组织已制定了 CA-125 进展标准,即将被加入到卵巢癌一线治疗方案的肿瘤客观评价标准中。

细胞学/组织学技术:在方案规定的特定情况下,这些技术可用于鉴定 PR 和 CR (如生殖细胞肿瘤的病灶中常存在残留的良性肿瘤组织)。当渗出可能是某种疗法潜在的副反应(如使用紫杉烷化合物或血管生成抑制剂的治疗),且可测量肿瘤符合缓解或疾病稳定标准时,在治疗过程中肿瘤相关的渗出出现或加重,可通过细胞学技术来确诊,以区分缓解(或疾病稳定)和疾病进展。

#### 2. 肿瘤缓解评估

### 2.1 全部肿瘤和可测量病灶的评估

为评价客观缓解或未来可能的进展,有必要对所有肿瘤病灶肿瘤的总负荷进行基线评估,为后面的测量结果作参照。在以客观缓解作为主要治疗终点的临床方案中,只有在基线时具有可测量病灶的受试者才能入选。可测量病灶定义为存在至少一处可测量的病灶。而对于那些以疾病进展(疾病进展时间或固定日期进展程度)为主要治疗终点的试验,方案入选标准中必须明确是仅限于有可测量病灶的受试者,还是没有可测量病灶也可以入选。

#### 2.2 靶病灶和非靶病灶的基线记录

基线评估时有超过一个以上可测量病灶时,应记录并测量所有病灶,总数不超过 5 个 (每个器官不超过 2 个),作为靶病灶代表所有累及器官(也就是说只有一个或两个累计器官的受试者最多选择两个或四个靶病灶作为基线测量病灶)。 靶病灶必须基于尺寸进行选择(最长直径),能代表所有累及器官,且测量必须具有良好的重复性。有时候当最大的病灶不能重复测量时可重新选择一个可重复测量的最大病灶。

淋巴结因其为正常组织且即使没有肿瘤转移仍可为影像察觉而需要特别关注。定义为可测量结节甚至是靶病灶的病理性淋巴结必须符合以下标准: CT 测量短直径≥15 mm。基线只需要检测短直径。放射学家通常借助结节的短直径来判断该结节是否已有肿瘤转移。结节尺寸一般用影像检测的两维数据来表示(CT 用轴平面,MRI 则从轴面、矢状面或冠状面中选择一个平面)。取最小值即为短直径。例如,一个 20 mm× 30 mm 的腹部结节短直径为 20 mm,可视为恶性的、 可测量的结节。在这个例子中,20mm 即是结节的测量值。直径≥10 mm 但<15 mm 的结节不应该视为靶病灶。而<10 mm 的结节则不属于病理结节范畴,不必予以记录和进一步观察。

所有靶病灶的直径经过计算所求之和(包括非结节病灶的最长直径和结节病灶的短直径) 将作为基线直径总和上报。如含有淋巴结直径,如上面提到的,只将短直径计算在内。基线 直径总和将作为疾病基线水平的参考数值。余所有的病灶包括病理淋巴结可视为非靶病灶, 无需进行测量,但应在基线评估时进行记录。如记录为"存在","缺失"或极少数情况下"明确进展"。广泛存在的靶病灶可与靶器官记录在一起(如大量扩增骨盆淋巴结或大规模肝转移)。

#### 2.3 缓解标准

#### 2.3.1 靶病灶评估

完全缓解(CR): 所有靶病灶消失,全部病理淋巴结(包括靶结节和非靶结节)短直径必须减少至<10 mm。

部分缓解 (PR): 靶病灶直径之和比基线水平减少至少 30%。

疾病进展(PD): 以整个实验研究过程中所有测量的靶病灶直径之和的最小值为参照,直径和相对增加至少 20%(如果基线测量值最小就以基线值为参照);除此之外,必须满足直径和的绝对值增加至少 5 mm(出现一个或多个新病灶也视为疾病进展)。

疾病稳定(SD): 靶病灶减小的程度没达到 PR,增加的程度也没达到 PD 水平,介于两者之间,研究时可以直径之和的最小值作为参考。

### 2.3.2 靶病灶评估的注意事项:

淋巴结:即使鉴定为靶病灶的淋巴结减小至 10 mm 以内,每次测量时仍需记录与基线对应的实际短直径的值(与基线测量时的解剖平面一致)这意味着如果淋巴结属于靶病灶,即使达到完全缓解的标准,也不能说病灶已全部消失, 因为正常淋巴结的短直径就定义为 <10 mm。在 CRF 表或其他的记录方式中需在特定位置专门记录靶淋巴节病灶;对于 CR,所有淋巴节短直径必须<10 mm; 对于 PR、SD 和 PD,靶淋巴节短直径实际测量值将被包含在靶病灶直径的和之中。

小到无法测量的靶病灶:临床研究中,基线记录过的所有病灶(结节或非结节)在后面的评估中都应再次记录实际测量值,即使病灶非常小(如2mm)。但有时候可能太小导致CT扫描出的图像十分模糊,放射科医生也很难定义出确切的数值,就可能报告为"太小而测量不到"。出现这种情况时,在CRF表上记录上一个数值是十分重要的。如果放射科医生认为病灶可能消失了,那也应该记录为0mm。如果病灶确实存在但比较模糊,无法给出精确的测量值时,可默认为5mm。(注:淋巴结出现这种情况的可能性不大,因其正常情况下一般都具有可测量的尺寸,或者像在腹膜后腔中一样常常为脂肪组织所包绕;但是如果也出现这种无法给出测量值的情况,也默认为5mm)。5mm的默认值源于CT扫描的切割厚度(这个值不因C不同的切割厚度值而改变)。由于同一测量值重复出现的几率不大,提供这个默认值将降低错误评估的风险。但需要重申的是,如果放射医生能给出病灶大小的确切数值,即使病灶直径小于5mm,也必须记录实际值。

分离或结合的病灶: 当非结节性病灶分裂成碎片状时,将各分离部分的最长径加起来计算病灶的直径之和。同样,对于结合型病灶,通过各结合部分间的平面可将其区分开来,然后计算各自的最大直径。但如果结合得密不可分,最长径应取融合病灶整体的最长径。

### 2.3.3 非靶病灶的评估

这部分对非靶病灶肿瘤的缓解标准进行了定义。虽然一些非靶病灶实际可测量,但无需测量,只需在方案规定的时间点进行定性评估即可。

完全缓解(CR): 所有非靶病灶消失,且肿瘤标记物恢复至正常水平。所有淋巴结为非病理尺寸(短径<10 mm)。

非完全缓解/非疾病进展:存在一个或多个非靶病灶和/或持续存在肿瘤标记物水平超出正常水平。

疾病进展:已存在的非靶病灶出现明确进展。注:出现一个或多个新病灶也被视为疾病进展。

#### 2.3.4 关于的非靶病灶进展评估的特别注意事项

关于非靶病灶进展的定义补充解释如下: 当受试者存在可测量非靶病灶时,即使靶病灶评估为稳定或部分缓解,要在非靶病灶的基础上作出明确进展的定义, 必须满足非靶病灶整体的恶化程度已达到必须终止治疗的程度。而一个或多个非靶病灶尺寸的一般性增大往往

不足以达到进展标准,因此,在靶病灶为稳定或部分缓解时,仅依靠非靶病灶的改变就能定义整体肿瘤进展的情况几乎是十分稀少的。当受试者的非靶病灶均不可测量时:在一些III期试验中,当入选标准中没有规定必须存在可测量病灶时,就会出现这种情况。整体评估还是参照上文标准,但因为这种情况下没有病灶的可测量数据。非靶病灶的恶化不容易评估(根据定义:必须所有非靶病灶都确实无法测量),因此当非靶病灶改变导致整体疾病负荷增加的程度相当于靶病灶出现疾病进展时,依据非靶病灶作出明确进展的定义,需要建立一种有效的检测方法来进行评估。如描述为肿瘤负荷增加相当于体积额外增加73%(相当于可测量病灶直径增加20%)。又比如腹膜渗出从"微量"到"大量";淋巴管病变从"局部"到"广泛播散";或在方案中描述为"足够至改变治疗方法"。例子包括胸膜渗出液从痕量到大量,淋巴受累从原发部位向远处扩散,或者在方案中可能被描述为"有必要进行治疗方面的改变"。如果发现有明确的进展,该受试者应该在那个时点总体上视为疾病进展。最好具有客观标准可适用于不可测量的病灶的评估,注意,增加的标准必须是可靠的。

#### 2.3.5 新病灶

新的恶性病灶的出现预示着疾病的进展;因此针对新病变的一些评价是非常重要的。目前没有针对影像学检测病灶的具体标准,然而一种新的病灶的发现应该是明确的。比如说,进展不能归因于影像学技术的不同,成像形态的改变,或者肿瘤以外的其它病变(如:一些所谓新的骨病灶仅仅是原病灶的治愈,或原病灶的复发)。当病人的基线病灶出现部分或完全反应时,这一点非常重要的,例如:一例肝脏病灶的坏死可能在 CT 报告上定为新的囊性病变,而其实不是。

在随访中已检测到的而在基线检查中未发现的病灶将视为新的病灶,并提示疾病进展。例如一个在基线检查中发现有内脏病灶的受试者,当他做 CT 或 MRI 的头颅检查时发现有转移灶,该受试者的颅内转移病灶将被视为疾病进展的依据,即使他在基线检查时并未做头颅检查。

如果一个新的病灶是不明确的,比如因其形态小所致,则需要进一步的治疗和随访评价以确认其是否是一个新的病灶。如果重复的检查证实其是一个新的病灶,那么疾病进展的时间应从其最初的发现的时间算起。

病灶进行 FDG-PET 评估一般需要额外的检测进行补充确认,FDG-PET 检查和补充 CT 检查结果相结合评价进展情况是合理的(尤其是新的可疑疾病)。新的病灶可通过 FDG-PET 检查予明确的,依据以下程序执行:

基线 FDG-PET 检查结果是阴性的,接下来随访的 FDG-PET 检查是阳性的,表明疾病的进展。 没有进行基线的 FDG-PET 检查,后续的 FDG-PET 检查结果是阳性的:如果随访的 FDG-PET 阳性检查结果发现的新的病变灶与经 CT 检查结果相符,证明是 疾病进展。

如果随访的 FDG-PET 的阳性检查结果发现的新的病变灶未能得到 CT 检查结果的确认,需再行 CT 检查予以确认(如果得到确认,疾病进展时间从前期 FDG-PET 检查发现异常算起)。

如果随访的 FDG-PET 的阳性检查结果与经 CT 检查已存在的病灶相符,而该病灶在影像学检测上无进展,则疾病无进展。

#### 2.4 最佳整体疗效评价

最佳整体疗效评价是从试验开始至试验结束的最佳疗效记录,同时要把任何必要条件考虑在内以便确认。有时疗效反应出现在治疗结束后,因此方案应该明确治疗结束后的疗效评价是否考虑在最佳整体疗效评价之内方案必须明确任何进展前新的治疗如何影响最佳疗效反应。受试者的最佳疗效反应主要依赖目标病灶和非目标病灶的结果以及新病灶的表现情况。此外,还依赖于试验性质、方案要求及结果衡量标准。具体来说,在非随机试验中,疗效反应情况是首要目标,PR 或 CR 的疗效确认是必须的,以确认哪个是最佳整体疗效反应。

#### 2.4.1 时间点反应

假设在每个方案的具体时间点上都会有疗效反应发生。 表 1 将提供一个基线水平上疾

病表可测量的受试者人群其在每个时间点上的总体疗效反应的总结。 如果受试者无可测量 病灶(无目标病灶),评估可参见表 2。

#### 2.4.2 评估缺失和不可评价说明

如果在某个特定时间点上无法进行病灶成像或测量,则该受试者在该时间点上无法评价。如果在一个评价中只能对部分病灶进行评价,通常这种情况视为在那个时间点无法评价,除非有证据证实缺失的病灶不会影响指定时间点的疗效反应评价。这种情况很可能发生在疾病进展的情况。例如:一个受试者在基线水平有3个总和为50mm的病灶,但是随后只有2个病灶可评价,总和为80mm,该受试者将被评价为疾病进展,不管缺失的病灶影响有多大。

### 2.4.3 最佳总缓解:全部时间点

一旦受试者的所有资料都具备,其最佳总缓解可以确定。

当研究不需要对完全或部分疗效反应进行确认时最佳总缓解的评估:试验中最佳疗效反应是所有时间点上的最佳反应(例如:一个受试者在第一周期疗效评价为 SD,第二周期评价为 PR,最后一周期评价为 PD,但其最佳总缓解评价为 PR。当最佳总缓解评价为 SD 时,其必须满足方案所规定的从基线水平算起的最短时间。如果没有达到最短时间的标准,即使最佳总缓解评价为 SD 也是不认可的,该受试者的最佳总缓解将视随后的评价而定。例如:一个受试者第一周期评价为 SD,第二周期为 PD,但其未达到 SD 的最短时间要求,其最佳总缓解评价为 PD。同样的受试者在第一周期评价为 SD 后失访将被视为不可评价。

当研究需要对完全或部分疗效反应进行确认时最佳总缓解的评估: 只有当每一个受试者符合试验规定的部分或者完全缓解标准而且在方案中特别提及的在随后的时间点(一般是四周后)再次做疗效确认后才能宣称是完全或者部分缓解。在这种情况下,最佳总缓解见表 3 的说明。

#### 2.4.4 疗效评估的特别提示

当结节性病灶被包括在总的靶病灶评估中,同时该结节大小缩小到"正常"大小时(<10 mm),它们依然会有一个病灶大小扫描报告。为了避免过高评估基于结节大小增加所反映的情况,即便是结节正常,测量结果也将被记录。正如前面已经提及的,这就意味着疗效为完全缓解的受试者,CRF表上也不会记录为0。

若试验过程中需要进行疗效确认,重复的"不可测量"时间点将使最佳疗效评估变得复杂。试验的分析计划必须说明,在确定疗效时,这些缺失的数据/评估可以被解释清楚。比如,在大部分试验中,可以将某受试者 PR-NE-PR 的反应作为得到了疗效确认。

当受试者出现健康情况整体恶化要求停止给药治疗,但是没有客观证据证明时,应该被报道为症状性进展。即便在治疗终止后也应该尽量去评估客观进展的情况。症状性恶化不是客观反应的评估描述:它是停止治疗的原因。那样的受试者的客观反应情况将通过表 1 到 3 所示的目标和非目标病灶情况进行评估。

定义为早期进展,早期死亡和不可评估的情况是研究特例,且应该在每个方案中进行明确的描述(取决于治疗间期和治疗周期)。

在一些情况下,从正常组织中辨别局部病灶比较困难。当完全缓解的的评估基于这样的定义时,我们推荐在进行局部病灶完全缓解的疗效评估前进行活检。 当一些受试者局部病灶影像学检测结果异常被认为是代表了病灶纤维化或者疤痕形成时,FDG-PET 被当作与活 检相似的评估标准,用来对完全缓解进行疗效确认。在此种情况下,应该在方案中对 FDG-PET 的应用进行前瞻性描述,同时以针对此情况专科医学文献的报告作为支持。但是必须意识到的是由于 FDG-PET 和活检本身的限制性(包括二者的分辨率和敏感性高低),将会导致完全缓解评估时的假阳性结果。

表 1. 时间点反应: 有靶病灶的受试者(包括或者不包括非靶病灶)

| 靶病灶 | 北脚岸体 | <b>杂</b> 化 | 总体缓解 |
|--------------|------|------------|------|
| 1 111777111. | 非靶病灶 | 新及伪江 | 尽体缓胀 |

| CR | CR | 非 | CR |
|---------|------------|---------|---------|
| CR | 非 CR/非 PD | 非 | PR |
| CR | 不能评估 | 非 | PR |
| PR | 非进展或不能完全评估 | 非 | PR |
| SD | 非进展或不能完全评估 | 非 | SD |
| 不能完全评估 | 非进展 | 非 | NE |
| PD | 任何情况 | 是或否 | PD |
| 任何情况 | PD | 是或否 | PD |
| 任何情况 | 任何情况 | 是 | PD |
| CR=完全缓解 | PR=部分缓解 | SD 疾病稳定 | PD=疾病进展 |
| | | | NE=不能评估 |

表 2. 时间点反应-仅有非目标病灶的受试者

| 非靶病灶 | 新发病灶 | 总体缓解 |
|-------------|------|-------------|
| CR | 非 | CR |
| 非 CR 或者非 PD | 非 | 非 CR 或者非 PD |
| 不能完全评估 | 非 | 不能评估 |
| 不能明确的 PD | 是或否 | PD |
| 任何情况 | 是 | PD |

注解:对于非目标病灶,"非 CR/非 PD"是指优于 SD 的疗效。由于 SD 越来越多作为评价疗效的终点指标,因而制定非 CR/非 PD 的疗效,以针对未规定无病灶可测量的情况。对于不明确的进展发现(如非常小的不确定的新病灶;原有病灶的囊性变或坏死病变)治疗可以持续到下一次评估。如果在下一次评估中,证实了疾病进展,进展日期应该是先前出现疑似进展的日期。

表 3. CR 和 PR 疗效需要确认的最佳总缓解

| 第一个时间点总 | 随后时间点总 | 最佳总体缓解 |
|---------|--------|----------------------------|
| 缓解 | 缓解 | |
| CR | CR | CR |
| CR | PR | SD,PD 或 PR <sup>a</sup> |
| CR | SD | 如果 SD 持续足够时间则为 SD, 否则应为 PD |
| CR | PD | 如果 SD 持续足够时间则为 SD, 否则应为 PD |
| CR | NE | 如果 SD 持续足够时间则为 SD, 否则应为 NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | 如果 SD 持续足够时间则为 SD, 否则应为 PD |
| PR | NE | 如果 SD 持续足够时间则为 SD, 否则应为 NE |
| NE | NE | NE |

注解: CR 即是完全缓解, PR 是部分缓解, SD 是疾病稳定, PD 是疾病进展, NE 即不可评价。上标"a": 如果在第一个时间点 CR 真正出现,在随后的时间点出现的任何疾病,那么即便相对于基线该受试者疗效达到 PR 标准,其疗效评价在之后的时间点仍然为 PD(因为在 CR 之后疾病将再次出现)。最佳缓解取决于是否在最短的治疗间隔内出现 SD。然而有时第一次

评价为 CR,但随后的时间点扫描提示小病灶似乎依然出现,因而实际上受试者疗效在第一个时间点应该是 PR 而不是 CR。在这种情况下,首次 CR 判断应该被修改为 PR,同时最好的反应是 PR。

#### 2.5. 肿瘤重新评价的频率

治疗期间肿瘤重新评价的频率决定于治疗方案,并应与治疗的类型和日程安排相符。但是在治疗的受益效果不清楚的II期试验中,每6~8周(时间设计在一个周期的结束点)进行随访是合理的,在特殊方案或情况下可调整时间间隔长度。方案应该具体指明哪些组织部位需要进行基线水平的评估(通常是那些最可能与所研究肿瘤类型的转移病变密切相关的组织部位)和评价重复的频率。正常情况下,靶病灶和非靶病灶在每次评估时都应进行评价,在一些可选择的情形下,某些非目标病灶评价频率可以小一些,例如,目标疾病的疗效评价确认为 CR 或怀疑有骨性病变进展时才需重复骨扫描。

治疗结束后,重新评价肿瘤取决于是否把缓解率或者是到出现某一事件(进展/死亡)的时间作为临床试验终点。如为出现某一事件时间(如 TTP/DFS/PFS)则需要进行方案中规定的常规重复评价。特别是在随机比较试验中预定的评价应该列在时间表内(如:治疗中的6~8周,或治疗后的3~4个月),不应受到其他因素的影响,如治疗延迟、给药间隔 和任何其他在疾病评价时间选择上可能导致治疗臂不均衡的事件等。

### 2.6. 疗效评估/缓解期的确认

### 2.6.1. 确认

对于以疗效为主要研究终点的非随机临床研究,必须对 PR 和 CR 的疗效进行确认,以保证疗效不是评价失误的结果。这也允许在有历史数据的情况下,对结果进行合理的解释,但这些试验的历史数据中的疗效也应进行过确认。但在所有其他情况下,如随机试验(II 或III期)或者以疾病稳定或者疾病进展为主要研究终点的研究中,不再需要疗效确认,因为这对于试验结果的解释没有价值。 然而取消疗效确认的要求,就会使防止偏移作用的中心审查 显得更加重要,特别是在非盲态实验研究中。

SD 的情况下,在试验开始后的最短时间间隔内(一般不少于 6~8 周),至少有一次测量符合方案中规定的 SD 标准。

#### 2.6.2 总缓解期

总缓解期是从测量首次符合 CR 或 PR (无论哪个先测量到)标准的时间到首次真实记录疾病复发或进展的时间(把试验中记录的最小测量值作为疾病进展的参考)。总完全缓解时间是从测量首次符合 CR 标准的时间到首次真实记录疾病复发或进展的时间。

### 2.6.3. 疾病稳定期

是从治疗开始到疾病进展的时间(在随机化试验中,从随机分组的时间开始),以试验中最小的总和作为参考(如果基线总和,最小则作 PD 计算的参考)。疾病稳定期的临床相关性因不同研究和不同疾病而不同。如果在某一特定的试验中,以维持最短时间稳定期的病人比例作为研究终点,方案应特别说明 SD 定义中两个测量间的最短时间间隔。

注意:缓解期、稳定期以及 PFS 受基线评价后随访频率的影响。定义标准随访频率不属于本指导原则范围。随访频率应考虑许多因素,如疾病类型和分期、治疗周期及标准规范等。但若需进行试验间的比较,应考虑这些测量终点准确度的限制。

#### **4.7. PFS/TTP**

### 4.7.1. II期临床试验

本指导原则主要关注II期临床试验中客观缓解作为研究终点的应用。在某些情况下,缓解率可能不是评价新药/新方案潜在抗癌活性的最优选择。在这些情况下,分界时间点上的PFS/PPF(Proportion progress-free,无进展比例)可认为是提供新药生物活性的原始信号的合适替代指标。但是很明显,在一个非对照试验中,这些评价会受到质疑,因为貌似有价值的观察可能与病人的筛选等生物学因素有关,而非药物干预的作用。因此,以这些作为研究终点的II期临床试验最好设计随机对照。但某些肿瘤的临床表现始终如一(通常一直状况

差) ,非随机试验也是合理的。但是在这些 情况下,因缺少阳性对照,评估预期 PFS 或 PPF 时,需小心记录疗效证据。

# 14. 附件二: ECOG 体力状况计分标准

# (东部肿瘤协作组)

| 计分 | 活动水平 |
|----|------------------------------------|
| 0 | 完全正常,能毫无限制地进行所有正常活动。 |
| 1 | 不能进行剧烈的体力活动,但可以走动,并能从事轻体力活动或办公室工作。 |
| 2 | 可以走动,生活可自理,但不能进行任何工作,白天卧床时间不超过50%。 |
| 3 | 生活勉强可以自理,白天超过50%的时间需要卧床或坐在椅子上休息。 |
| 4 | 完全丧失活动能力,生活严重不能自理,必须卧床或使用轮椅。 |
| 5 | 死亡。 |

# 15. 附件三: 纽约心脏病学会心功能分级(NYHA)

# 纽约心脏病学会心功能分级(NYHA)

| 级别 | 体力活动 | 症状(疲劳、心悸 | 季、气喘或心绞痛) | 静息状态 |
|-----|------|----------|-----------|--------------|
| I | 不受限 | 无症状 | 一般体力活 | 动不引起 |
| II | 轻度受限 | 无症状 | 日常体力活 | <b></b> 动可引起 |
| III | 明显受限 | 无症状 | 低于日常作 | 本力活动引起 |
| IV | 丧失 | 有症状 | 任何体力 | 舌动均加重 |

# 16. 附件四. 索凡替尼与伴随用药潜在相互作用的指导原则

目前还没有数据表明在有药代动力学方面索凡替尼和一些伴随用药之间有互相作用。

根据体外肝微粒体温孵试验中发现介导索凡替尼代谢的I相代谢酶主要有 CYP3A4/5 和 CYP2C8(脱氢、N-去甲基)、CYP2E1(单氧化)和 FMO。索凡替尼对 P450 酶无明显的抑制作用。在人原代肝细胞中对 CYP1A2 和 CYP3A 的诱导实验结果显示,索凡替尼在  $10\,\mu$ M 浓度下对 CYP1A2 和  $2\,\mu$ M 浓度下对 CYP3A4 不具有明显诱导作用。利用 Caco-2 细胞进行的通透性和外排转运的体外试验提示索凡替尼可能为外排转运体 P-gp 的底物。

根据体外试验, 索凡替尼对代谢酶 CYP3A4/5 有时间依赖性抑制作用, k<sub>inact</sub> 为 0.73 min<sup>-1</sup>, KI 为 163 μM。此附件中表 1-3 提供了一系列 CYP3A4 的强诱导剂、强抑制剂和底物。 受试者在接受第一剂试验药物治疗之前 3 周内接受贯叶连翘治疗或 2 周内接受过其他 CYP3A4 的强诱导剂或强抑制剂将不能参与这项研究。

试验过程中应该尽量避免同时使用 CYP3A4 的强诱导剂、强抑制剂或底物,除非由研究者认为是必须需要使用的,但在这种情况下,必须密切监测病人由于药物相互作用导致的试验药物疗效的降低或毒性的增加。

这些列表能够罗列的内容是有限的,其它已知的对 CYP3A4 活性有较强调节的药物、或主要由 CYP3A4 代谢的药物也应采取类似的限制。如有必要,在联合服用索凡替尼前,需参考所有联用药物的完整处方信息。

### 表 1. CYP3A4 酶抑制性较强的药物

可能增加索凡替尼暴露的 CYP3A4 的强抑制剂

波西普韦
克拉霉素
考尼伐坦
埃替格韦/利托那韦
氟康唑
葡萄柚汁 ab

茚地那韦
依曲康唑

酮康唑
洛匹那韦/利托那韦
米贝拉地尔
奈非那韦
泊沙康唑
利托那韦
沙奎那韦
特拉匹韦
泰利霉素
替拉那韦
利托那韦

### RIT = Ritonavir.利托那韦

a 高浓度的葡萄柚汁

伏立康唑

b 在参与研究期间,病人不应大量食用西柚和酸橙(以及其他含有这类水果的产品,例如西柚汁或者橘子酱),每天不应超过一小杯(120ml)西柚汁或者半个西柚,或者 1-2 勺(15g)橘子酱。

### 表 2 CVP3A4 酶的强诱导剂

| 衣 2. CYP3A4 瞬的独防守剂 |
|--------------------|
| CYP3A4 酶的强诱导剂 |
| 阿伐麦布 |
| 立痛定 |
| 恩杂鲁胺 |
| 米托坦 |
| 苯巴比妥米那 |
| 苯妥英 |
| 利福布 |
| 利福平 |
| 贯叶连翘 |
| 47 |

### 表 3 CYP3A4 酶的底物

| <b>₹3 CYP3A4 酶的底物</b> CYP3A4 酶的底物 |
|-----------------------------------|
| 阿瑞吡坦 |
| 布地缩松 |
| 丁螺环酮 |
| 考尼伐坦 |
| 达非那新 |
| 达芦那韦 |
| 达沙替尼 |
| 决奈达隆 |
| 依立曲坦 |
| 依普利酮 |
| 依维莫司 |
| 非洛地平 |
| 印地那韦 |
| 氟替卡松 |
| 洛匹那韦 |
| 洛伐他丁 |
| 鲁拉西酮 |
| 马拉维若 |
| 咪达唑仑 |
| 尼索地平 |
| 喹硫平 |
| 沙奎那韦 |
| 西地那非 |
| 辛伐他汀 |
| 西罗莫司 |
| 托伐普坦 |

| 替拉那韦 |
|-------|
| 三唑仑 |
| 替格瑞洛 |
| 伐地那非 |
| 阿司咪唑 |
| 西沙必利 |
| 环孢霉素 |
| 双氢麦角胺 |
| 麦角胺 |
| 芬太尼 |
| 哌迷清 |
| 奎尼丁 |
| 他克莫司 |
| 特非那定 |